CLINICAL TRIAL: NCT03000439
Title: EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF TOFACITINIB FOR TREATMENT OF SYSTEMIC JUVENILE IDIOPATHIC ARTHRITIS (SJIA) WITH ACTIVE SYSTEMIC FEATURES IN CHILDREN AND ADOLESCENT SUBJECTS
Brief Title: A Safety, Efficacy And Pharmacokinetics Study Of Tofacitinib In Pediatric Patients With sJIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921165; 2017-002018-29 (EudraCT Number)
Record Dates: First submitted 2016-11-09; First posted 2016-12-22 (Estimated); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Arthritis Juvenile Idiopathic
Keywords: systemic Juvenile Idiopathic Arthritis; Xeljanz; Tofacitinib; sJIA; CP-690 550
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tofacitinib 5 mg BID (Experimental): oral, twice daily, tablet or solution.
  Interventions: Drug: In open-label phase: treatment with tofacitinib; Drug: In double-blind phase: treatment with tofacitinib or placebo in 1:1 ratio
- Placebo (Placebo Comparator)
  Interventions: Drug: In double-blind phase: treatment with tofacitinib or placebo in 1:1 ratio

INTERVENTIONS:
Drug: In open-label phase: treatment with tofacitinib — Treatment with investigational drug
  Other Names: CP-690,550; Xeljanz
  Arms: Tofacitinib 5 mg BID
Drug: In double-blind phase: treatment with tofacitinib or placebo in 1:1 ratio — Treatment with investigational drug or placebo
  Other Names: CP-690,550; Xeljanz

SUMMARY:
A randomized withdrawal study in which responders to open-label treatment with tofacitinib will be randomized in a 1:1 ratio to tofacitinib or placebo in a double-blind phase. In the double-blind phase "time to sJIA flare" will be evaluated as primary endpoint and subjects will be discontinued once they experience sJIA flare. An interim analysis for efficacy and futility will be conducted when at least 20 flares have been observed. If either criterion is met, the study will be stopped. If neither criterion is met, the study will continue until the requisite number of flares are observed as determined by the number of flares included in the interim analysis and a statistical penalty for conducting the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* active sJIA disease according to ILAR criteria before screening and at baseline (Day 1);
* Treatment with stable doses of methotrexate (MTX) ≤25 mg/week or ≤20 mg/m2/week, whichever is lower, is permitted;
* Treatment with a stable dose of oral prednisone ≤1 mg/kg/day up to a maximum of 30 mg/day, or equivalent, for at least 1 week before the first study drug dose is permitted.

Exclusion Criteria:

* Previous juvenile idiopathic arthritis (JIA) treatment with tofacitinib.
* Current symptoms or findings of myocarditis, endocarditis or more than minimal pericardial effusion associated with systemic juvenile idiopathic arthritis (sJIA). Current symptoms or findings of more than minimal pleuritis with sJIA.
* Current infection or serious infection within 3 months of study enrollment.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cohen Children's Medical Center of New York, Lake Success, New York
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
- Argentina (2):
  - Instituto CAICI SRL, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Brazil (4):
  - Faculdade de Medicina da UNESP, Botucatu, São Paulo
  - UPECLIN Unidade de Pesquisa Clinica da Faculdade de Medicina da UNESP, Botucatu, São Paulo
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina, São Paulo
  - Instituto da Crianca do Hospital das Clinicas da FMUSP, São Paulo
- Canada (2):
  - Alberta Children's Hospital/University of Calgary, Calgary, Alberta
  - Research Institute of McGill University Health Center, Glen site, Montreal, Quebec
- China (9):
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Xi'an Children's Hospital, Xi'an, Shaanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - The Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Children's Hospital, Capital Medical University/Rheumatology Department, Beijing
- Hospital Metropolitano, San José, Costa Rica
- Germany (2):
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - St. Josef-Stift Sendenhorst, Sendenhorst
- Semmelweis Egyetem, Budapest, Hungary
- India (4):
  - Nirmal Hospital Pvt Ltd, Surat, Gujarat
  - Sir Ganga Ram Hospital, Rajinder Nagar, NEW Delhi
  - Institute of Child Health, Kolkata, West Bengal
  - Institute of Post Graduate Medical Education and Research & SSKM Hospital, Kolkata, West Bengal
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center - Pediatric Clinic, Kfar Saba
- Italy (2):
  - Istituto Giannina Gaslini Istituto Pediatrico di Ricovero e Cura a Carattere Scientifico, Genova, Genoa
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milan
- Mexico (3):
  - Clínica de Investigacion en Reumatologia y Obesidad, S.C., Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi, S.C., San Luis Potosí City
- Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw, Poland
- Russia (2):
  - Clinic of FSBEI HE BSMU MoH RF, Ufa, Bashkortostan Republic
  - Federal State Budgetary Scientific Institution "Scientific and Research Rheumatology, Moscow
- South Africa (2):
  - Enhancing Care Foundation, Durban, KwaZulu-Natal
  - Panorama Medical Centre, Cape Town, Western Cape
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital Department of Pediatric Rheumatology, Kadikoy / Istanbul
- Ukraine (4):
  - Communal Institution "Dnipropetrovsk Specialized Clinical Medical Center of Mother and Child n.a., Dnipro
  - Municipal non-Profit Enterprise, Ivano-Frankivsk
  - CNE of Lviv Regional Council "Western Ukrainian Specialized Pediatric, Lviv
  - Vinnytsia Regional Children's Clinical Hospital, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were diagnosed with Systemic Juvenile Idiopathic Arthritis (sJIA) with active systemic features were enrolled.
Pre-assignment Details: A total of 168 participants were screened, of which 68 failed screening and only 100 participants were enrolled in open label part 1 (OLP1). From the total of 100 participants enrolled into OLP1 of the study, 54 participants were treated in open label part 2 (OLP2), and 59 participants were randomized between the treatment groups in the double-blinded (DB) phase.
Groups:
- Tofacitinib 5mg BID Open-Label (OL) Part 1: Participants were administered tofacitinib 5 milligram (mg) twice a day (BID) via the oral route and continued to receive a stable dose of corticosteroids (Cs) during open label part 1.
- Tofacitinib 5mg BID OL Part 2: Participants who achieved sJIA American college of rheumatology (ACR) 50 response and maintained sJIA ACR 30 response for 4 weeks were administered tofacitinib 5 mg BID and tapering dose of CSs for participants treated with greater than (˃0.2) milligram/kilogram/day (mg/kg/day) oral prednisone (or equivalent).
- Tofacitinib 5mg BID DB: Participants who maintained a stable tapered CS dose for 4 weeks and maintained sJIA ACR 30 for 4 weeks from Part 1 and Part 2 of the open-label phase continued to receive tofacitinib 5 mg BID orally during the double-blind withdrawal phase of the study.
- Placebo DB: Participants who maintained a stable tapered CS dose for 4 weeks and maintained sJIA ACR 30 for 4 weeks from Part 1 and Part 2 of the open-label phase were randomized to receive placebo BID orally during the double-blind withdrawal phase of the study.
Period: Open Label Part 1
Arm/Group | Tofacitinib 5mg BID Open-Label (OL) Part 1 | Tofacitinib 5mg BID OL Part 2 | Tofacitinib 5mg BID DB | Placebo DB
Started | 100 | 0 | 0 | 0
Completed | 76 | 0 | 0 | 0
Not Completed | 24 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0
Not completed — Insufficient clinical response | 16 | 0 | 0 | 0
Period: Open Label Part 2
Arm/Group | Tofacitinib 5mg BID Open-Label (OL) Part 1 | Tofacitinib 5mg BID OL Part 2 | Tofacitinib 5mg BID DB | Placebo DB
Started | 0 | 54 | 0 | 0
Completed | 0 | 37 | 0 | 0
Not Completed | 0 | 17 | 0 | 0
Not completed — Other | 0 | 5 | 0 | 0
Not completed — Insufficient clinical response | 0 | 12 | 0 | 0
Period: Double Blind Phase
Arm/Group | Tofacitinib 5mg BID Open-Label (OL) Part 1 | Tofacitinib 5mg BID OL Part 2 | Tofacitinib 5mg BID DB | Placebo DB
Started | 0 | 0 | 28 | 31
Completed | 0 | 0 | 14 | 17
Not Completed | 0 | 0 | 14 | 14
Not completed — Adverse Event | 0 | 0 | 2 | 1
Not completed — Withdrawal by parent/guardian | 0 | 0 | 2 | 0
Not completed — Other | 0 | 0 | 10 | 11
Not completed — Insufficient clinical response | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall: All participants who received at least one dose of investigational product in the study.
Arm/Group | Overall
Number analyzed (Participants) | 100
Age, Customized [Count of Participants; unit: Participants]
  2 to less than (<) 6 Years | 17
  6 to < 12 Years | 43
  12 to < 18 Years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 39
  Race: Black or African American | 7
  Race: Asian | 49
  Race: Other | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 14
  Ethnicity: Not Hispanic or Latino | 86

OUTCOME MEASURES:

1. Primary Outcome: Time to Systemic Juvenile Idiopathic Arthritis (sJIA) Disease Flare: Double-Blind Phase
Description: Time to the disease flare=the number of days from randomization to flare in the DB phase and calculated as date of disease flare minus (-) date of randomization plus (+) 1. sJIA Flare=as at least one of the following criteria: Recurrence of fever >38 degree Celsius (C)/100.4 degree Fahrenheit (F) on 2 or more consecutive days) was considered due to SJIA activity. Worsening of 30 percent (%) or more in three or more of the six variables included: Number of joints with active arthritis and limited range of motion, disease activity, parent child evaluation of overall well-being, functional ability, childhood health assessment questionnaire ( CHAQ disability index), erythrocyte sedimentation rate (ESR) millimeter/ hour (mm/hr), of the JIA core set with no more than one variable of the JIA core set improving by 30% compared to the day of randomization into the withdrawal phase. 95% Confidence Interval (CI) based on Brookmeyer and Crowley Method.
Time Frame: From randomization up to 248 weeks
Population: Double blind full analysis set (DBFAS) consisted of all randomized participants who received at least one dose of investigational product in the DB phase.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Tofacitinib 5mg BID DB: Participants who maintained a stable tapered CS dose for 4 weeks and maintained sJIA ACR 30 for 4 weeks from Part 1 and Part 2 of the OL phase continued to receive tofacitinib 5 mg BID orally during the DB withdrawal phase of the study.
- Placebo DB: Participants who maintained a stable tapered CS dose for 4 weeks and maintained sJIA ACR 30 for 4 weeks from Part 1 and Part 2 of the OL phase were randomized to receive placebo BID orally during the DB withdrawal phase of the study.
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Days | NA [186.0 to NA] — Median and upper limit of 95% CI were not estimated due to insufficient number of participants with event. | 295.0 [99.0 to NA] — Upper limit of 95% CI was not estimated due to insufficient number of participants with event.
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; Test type: Other; p = 0.1171, Unstratified log-rank test — 1-sided p-value is provided; Hazard Ratio (HR) = 0.633, 95% CI 2-sided [0.296 to 1.354] — Hazard ratio and 95% CI was based on Cox proportional hazards model with treatment group as covariate. Hazard ratio < 1 indicates a reduction in hazard ratio in favor of Tofacitinib 5 mg BID to Placebo

2. Secondary Outcome: Probability of Occurrence of sJIA Disease Flare at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52: Double-Blind Phase
Description: sJIA Flare was defined as at least one of the following criteria: recurrence of fever (>38° C/100.4 degree F) on 2 or more consecutive days) was considered due to SJIA activity. Worsening of 30% or more in three or more of the six variables: number of joints with active arthritis and limited range of motion, disease activity, parent child evaluation of overall well-being, functional ability (CHAQ Disability Index), ESR. of the JIA core set with no more than one variable of the JIA core set improving by 30% compared to the day of randomization into the withdrawal phase. Probability of occurrence of sJIA disease flare with 95% CI were estimated using Kaplan-Meier method and reported in this outcome measure.
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: DBFAS consisted of all randomized participants who received at least one dose of investigational product in the DB phase.
Measure: Number; unit: Percentage probability of occurrence
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage probability of occurrence
  DB Week 4 | 7.1 | 6.5
  DB Week 8 | 14.3 | 22.6
  DB Week 12 | 21.4 | 32.3
  DB Week 16 | 25.0 | 38.7
  DB Week 20 | 32.1 | 45.4
  DB Week 24 | 32.1 | 45.4
  DB Week 28 | 35.9 | 45.4
  DB Week 32 | 35.9 | 49.9
  DB Week 36 | 40.5 | 49.9
  DB Week 40 | 40.5 | 49.9
  DB Week 44 | 40.5 | 55.5
  DB Week 48 | 40.5 | 55.5
  DB Week 52 | 40.5 | 55.5
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4; Test type: Other; Difference in percentage = 0.7, 95% CI 2-sided [-12.2 to 13.6] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8; Test type: Other; Difference in percentage = -8.3, 95% CI 2-sided [-27.9 to 11.3] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12; Test type: Other; Difference in percentage = -10.8, 95% CI 2-sided [-33.2 to 11.6] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16; Test type: Other; Difference in percentage = -13.7, 95% CI 2-sided [-37.2 to 9.8] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20; Test type: Other; Difference in percentage = -13.2, 95% CI 2-sided [-37.9 to 11.5] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24; Test type: Other; Difference in percentage = -13.2, 95% CI 2-sided [-37.9 to 11.5] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28; Test type: Other; Difference in percentage = -9.4, 95% CI 2-sided [-34.5 to 15.6] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32; Test type: Other; Difference in percentage = -14.0, 95% CI 2-sided [-39.5 to 11.5] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36; Test type: Other; Difference in percentage = -9.4, 95% CI 2-sided [-35.5 to 16.7] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40; Test type: Other; Difference in percentage = -9.4, 95% CI 2-sided [-35.5 to 16.7] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44; Test type: Other; Difference in percentage = -15.0, 95% CI 2-sided [-41.8 to 11.8] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48; Test type: Other; Difference in percentage = -15.0, 95% CI 2-sided [-41.8 to 11.8] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52; Test type: Other; Difference in percentage = -15.0, 95% CI 2-sided [-41.8 to 11.8] — The 95% CIs for the differences between the treatment groups were generated using Greenwood's formula

3. Secondary Outcome: Percentage of Participants Who Achieved Successful Corticosteroid Tapering: at the End of Open-label Phase Part 2
Description: A successfully tapered participant was considered as the one that completed part 2 of the OL by reaching their target corticosteroid dose and maintained an adapted JIA American College of Rheumatology (ACR) 30 response for four weeks on this dose. The target CS dose at the end of part 2 included less than equal to (<=) 0.5 milligram/kilogram/day (mg/kg/day) up to a maximum dose of 15 milligram/ day (mg/day) oral prednisone (or equivalent) for CS>0.8 mg/kg/day oral prednisone; reduction to <=0.3 mg/kg/day up to a maximum of 12 mg/day oral prednisone (or equivalent) for CS <=0.8 mg/kg/day to greater than equal to (>=) 0.5 mg/kg/day oral prednisone (or equivalent) and <=0.2 mg/kg/day up to a maximum dose of 10 mg/day oral prednisone (or equivalent) for CS <0.5 mg/kg/day-CS˃0.2 mg/kg/day oral prednisone (or equivalent). 95% CI was based on normal approximation.
Time Frame: From end of OL Part 1 to up to 24 weeks in OL Part 2
Population: Open-label part 2 (OLP2) analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tofacitinib 5mg BID OL Part 2: Participants who achieved sJIA ACR 50 response and maintained sJIA ACR 30 response for 4 weeks were administered tofacitinib 5 mg BID and tapering dose of CSs for participants treated with >0.2 mg/kg/day oral prednisone (or equivalent).
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants | 70.37 [58.19 to 82.55]

4. Secondary Outcome: Percentage of Participants Who Achieved Corticosteroid Dose of <= 0.2 mg/kg/Day or 10 mg/Day: at the End of Open-label Phase Part 2
Description: 95% CI was based on normal approximation.
Time Frame: From end of OL Part 1 to up to 24 weeks in OL Part 2
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants | 59.26 [46.15 to 72.36]

5. Secondary Outcome: Percentage of Participants With Adapted JIA ACR 30/50/70/90/100 Response at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: Adapted JIA ACR 30,50,70,90,100 response=absence of fever due to sJIA in preceding 7 days along with improvement of >=30,50,70,90,100%, respectively in at least 3 out of 6 JIA core set variables with no more than 1 JIA core set variable worsening by >=30%.Variables included: number of joints with active arthritis(any joint with swelling, or absence of swelling, limitation of motion accompanied by either pain on motion or tenderness);number of joints with limited range of motion; physician global evaluation of disease activity on VAS from 0=no disease activity to 10=very severe disease activity, higher scores:greater disease activity; parent/legal guardian/child evaluation of overall well-being on VAS from 0=very well to 10mm=very poor, higher scores: worsen condition; functional ability (Disability Index ranged from 0=no or minimal physical dysfunction, 3=very severe physical dysfunction, higher scores:more physical dysfunction;ESR (mm/hr).Missing response was imputed as non-response.
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage of participants
  ACR30:DB Week 4 | 82.14 [67.96 to 96.33] | 93.55 [84.90 to 100]
  ACR30:DB Week 8 | 82.14 [67.96 to 96.33] | 80.65 [66.74 to 94.55]
  ACR30:DB Week 12 | 71.43 [54.70 to 88.16] | 70.97 [54.99 to 86.95]
  ACR30:DB Week 16 | 71.43 [54.70 to 88.16] | 61.29 [44.14 to 78.44]
  ACR30:DB Week 20 | 67.86 [50.56 to 85.16] | 51.61 [34.02 to 69.21]
  ACR30:DB Week 24 | 64.29 [46.54 to 82.03] | 54.84 [37.32 to 72.36]
  ACR30:DB Week 28 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR30:DB Week 32 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR30:DB Week 36 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR30:DB Week 40 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR30:DB Week 44 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR30:DB Week 48 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR30:DB Week 52 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR50:DB Week 4 | 82.14 [67.96 to 96.33] | 93.55 [84.90 to 100]
  ACR50:DB Week 8 | 82.14 [67.96 to 96.33] | 77.42 [62.70 to 92.14]
  ACR50:DB Week 12 | 71.43 [54.70 to 88.16] | 70.97 [54.99 to 86.95]
  ACR50:DB Week 16 | 71.43 [54.70 to 88.16] | 58.06 [40.69 to 75.44]
  ACR50:DB Week 20 | 67.86 [50.56 to 85.16] | 48.39 [30.79 to 65.98]
  ACR50:DB Week 24 | 64.29 [46.54 to 82.03] | 54.84 [37.32 to 72.36]
  ACR50:DB Week 28 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR50:DB Week 32 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR50:DB Week 36 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR50:DB Week 40 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR50:DB Week 44 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR50:DB Week 48 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR50:DB Week 52 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR70:DB Week 4 | 57.14 [38.81 to 75.47] | 70.97 [54.99 to 86.95]
  ACR70:DB Week 8 | 67.86 [50.56 to 85.16] | 77.42 [62.70 to 92.14]
  ACR70:DB Week 12 | 64.29 [46.54 to 82.03] | 64.52 [47.67 to 81.36]
  ACR70:DB Week 16 | 60.71 [42.62 to 78.80] | 54.84 [37.32 to 72.36]
  ACR70:DB Week 20 | 64.29 [46.54 to 82.03] | 45.16 [27.64 to 62.68]
  ACR70:DB Week 24 | 53.57 [35.10 to 72.04] | 51.61 [34.02 to 69.21]
  ACR70:DB Week 28 | 57.14 [38.81 to 75.47] | 41.94 [24.56 to 59.31]
  ACR70:DB Week 32 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR70:DB Week 36 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  ACR70:DB Week 40 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR70:DB Week 44 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR70:DB Week 48 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR70:DB Week 52 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  ACR90:DB Week 4 | 28.57 [11.84 to 45.30] | 48.39 [30.79 to 65.98]
  ACR90:DB Week 8 | 21.43 [6.23 to 36.63] | 38.71 [21.56 to 55.86]
  ACR90:DB Week 12 | 25.00 [8.96 to 41.04] | 38.71 [21.56 to 55.86]
  ACR90:DB Week 16 | 25.00 [8.96 to 41.04] | 29.03 [13.05 to 45.01]
  ACR90:DB Week 20 | 21.43 [6.23 to 36.63] | 29.03 [13.05 to 45.01]
  ACR90:DB Week 24 | 21.43 [6.23 to 36.63] | 25.81 [10.40 to 41.21]
  ACR90:DB Week 28 | 17.86 [3.67 to 32.04] | 25.81 [10.40 to 41.21]
  ACR90:DB Week 32 | 14.29 [1.32 to 27.25] | 29.03 [13.05 to 45.01]
  ACR90:DB Week 36 | 28.57 [11.84 to 45.30] | 35.48 [18.64 to 52.33]
  ACR90:DB Week 40 | 28.57 [11.84 to 45.30] | 32.26 [15.80 to 48.71]
  ACR90:DB Week 44 | 28.57 [11.84 to 45.30] | 29.03 [13.05 to 45.01]
  ACR90:DB Week 48 | 28.57 [11.84 to 45.30] | 29.03 [13.05 to 45.01]
  ACR90:DB Week 52 | 28.57 [11.84 to 45.30] | 29.03 [13.05 to 45.01]
  ACR100:DB Week 4 | 14.29 [1.32 to 27.25] | 35.48 [18.64 to 52.33]
  ACR100:DB Week 8 | 10.71 [0 to 22.17] | 29.03 [13.05 to 45.01]
  ACR100:DB Week 12 | 14.29 [1.32 to 27.25] | 25.81 [10.40 to 41.21]
  ACR100:DB Week 16 | 17.86 [3.67 to 32.04] | 25.81 [10.40 to 41.21]
  ACR100:DB Week 20 | 14.29 [1.32 to 27.25] | 12.90 [1.10 to 24.70]
  ACR100:DB Week 24 | 17.86 [3.67 to 32.04] | 19.35 [5.45 to 33.26]
  ACR100:DB Week 28 | 14.29 [1.32 to 27.25] | 22.58 [7.86 to 37.30]
  ACR100:DB Week 32 | 10.71 [0 to 22.17] | 25.81 [10.40 to 41.21]
  ACR100:DB Week 36 | 14.29 [1.32 to 27.25] | 25.81 [10.40 to 41.21]
  ACR100:DB Week 40 | 21.43 [6.23 to 36.63] | 29.03 [13.05 to 45.01]
  ACR100:DB Week 44 | 21.43 [6.23 to 36.63] | 25.81 [10.40 to 41.21]
  ACR100:DB Week 48 | 25.00 [8.96 to 41.04] | 25.81 [10.40 to 41.21]
  ACR100:DB Week 52 | 25.00 [8.96 to 41.04] | 25.81 [10.40 to 41.21]
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 4; Test type: Other; Difference in percentage = -11.41, 95% CI 2-sided [-28.02 to 5.21] — The normal approximation to the difference in binomial proportions was used to generate 95% CI for the difference in percentage
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 8; Test type: Other; Difference in percentage = 1.50, 95% CI 2-sided [-18.37 to 21.36] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 12; Test type: Other; Difference in percentage = 0.46, 95% CI 2-sided [-22.68 to 23.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 16; Test type: Other; Difference in percentage = 10.14, 95% CI 2-sided [-13.82 to 34.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 20; Test type: Other; Difference in percentage = 16.24, 95% CI 2-sided [-8.43 to 40.92] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 24; Test type: Other; Difference in percentage = 9.45, 95% CI 2-sided [-15.49 to 34.39] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 28; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 32; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 36; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 40; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 44; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 48; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR30 at DB Week 52; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 14: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 4; Test type: Other; Difference in percentage = -11.41, 95% CI 2-sided [-28.02 to 5.21] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 15: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 8; Test type: Other; Difference in percentage = 4.72, 95% CI 2-sided [-15.72 to 25.17] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 16: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 12; Test type: Other; Difference in percentage = 0.46, 95% CI 2-sided [-22.68 to 23.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 17: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 16; Test type: Other; Difference in percentage = 13.36, 95% CI 2-sided [-10.76 to 37.48] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 18: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 20; Test type: Other; Difference in percentage = 19.47, 95% CI 2-sided [-5.20 to 44.14] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 19: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 24; Test type: Other; Difference in percentage = 9.45, 95% CI 2-sided [-15.49 to 34.39] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 20: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 28; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 21: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 32; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 22: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 36; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 23: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 40; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 24: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 44; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 25: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 48; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 26: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR50 at DB Week 52; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 27: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 4; Test type: Other; Difference in percentage = -13.82, 95% CI 2-sided [-38.14 to 10.49] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 28: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 8; Test type: Other; Difference in percentage = -9.56, 95% CI 2-sided [-32.28 to 13.15] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 29: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 12; Test type: Other; Difference in percentage = -0.23, 95% CI 2-sided [-24.70 to 24.24] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 30: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 16; Test type: Other; Difference in percentage = 5.88, 95% CI 2-sided [-19.31 to 31.06] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 31: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 20; Test type: Other; Difference in percentage = 19.12, 95% CI 2-sided [-5.81 to 44.06] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 32: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 24; Test type: Other; Difference in percentage = 1.96, 95% CI 2-sided [-23.55 to 27.47] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 33: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 28; Test type: Other — The normal approximation to the difference in binomial proportions was used to generate 95% CI for the difference in percentage; Difference in percentage = 15.21, 95% CI 2-sided [-10.05 to 40.46] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 34: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 32; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 35: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 36; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 36: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 40; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 37: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 44; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 38: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 48; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 39: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR70 at DB Week 52; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 40: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 4; Test type: Other; Difference in percentage = -19.82, 95% CI 2-sided [-44.09 to 4.46] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 41: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 8; Test type: Other; Difference in percentage = -17.28, 95% CI 2-sided [-40.19 to 5.63] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 42: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 20; Test type: Other; Difference in percentage = -7.60, 95% CI 2-sided [-29.66 to 14.45] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 43: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 12; Test type: Other; Difference in percentage = -13.71, 95% CI 2-sided [-37.19 to 9.77] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 44: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 16; Test type: Other; Difference in percentage = -4.03, 95% CI 2-sided [-26.67 to 18.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 45: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 32; Test type: Other; Difference in percentage = -14.75, 95% CI 2-sided [-35.32 to 5.83] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 46: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 24; Test type: Other; Difference in percentage = -4.38, 95% CI 2-sided [-26.02 to 17.26] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 47: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 28; Test type: Other; Difference in percentage = -7.95, 95% CI 2-sided [-28.89 to 12.99] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 48: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 36; Test type: Other; Difference in percentage = -6.91, 95% CI 2-sided [-30.65 to 16.83] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 49: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 40; Test type: Other; Difference in percentage = -3.69, 95% CI 2-sided [-27.16 to 19.78] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 50: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 44; Test type: Other; Difference in percentage = -0.46, 95% CI 2-sided [-23.60 to 22.68] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 51: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 48; Test type: Other; Difference in percentage = -0.46, 95% CI 2-sided [-23.60 to 22.68] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 52: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR90 at DB Week 52; Test type: Other; Difference in percentage = -0.46, 95% CI 2-sided [-23.60 to 22.68] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 53: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 4; Test type: Other; Difference in percentage = -21.20, 95% CI 2-sided [-42.45 to 0.05] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 54: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 8; Test type: Other; Difference in percentage = -18.32, 95% CI 2-sided [-37.98 to 1.34] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 55: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 12; Test type: Other; Difference in percentage = -11.52, 95% CI 2-sided [-31.65 to 8.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 56: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 16; Test type: Other; Difference in percentage = -7.95, 95% CI 2-sided [-28.89 to 12.99] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 57: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 20; Test type: Other; Difference in percentage = 1.38, 95% CI 2-sided [-16.15 to 18.91] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 58: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 24; Test type: Other; Difference in percentage = -1.50, 95% CI 2-sided [-21.36 to 18.37] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 59: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 28; Test type: Other; Difference in percentage = -8.29, 95% CI 2-sided [-27.91 to 11.32] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 60: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 32; Test type: Other; Difference in percentage = -15.09, 95% CI 2-sided [-34.29 to 4.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 61: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 36; Test type: Other; Difference in percentage = -11.52, 95% CI 2-sided [-31.65 to 8.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 62: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 40; Test type: Other; Difference in percentage = -7.60, 95% CI 2-sided [-29.66 to 14.45] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 63: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 44; Test type: Other; Difference in percentage = -4.38, 95% CI 2-sided [-26.02 to 17.26] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 64: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 48; Test type: Other; Difference in percentage = -0.81, 95% CI 2-sided [-23.04 to 21.43] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 65: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; ACR100 at DB Week 52; Test type: Other; Difference in percentage = -0.81, 95% CI 2-sided [-23.04 to 21.43] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants With Adapted JIA American College of Rheumatology (ACR) 30/50/70/90/100 Response at Part 1 Day 7, Weeks 2, 4, 8, 12, and 16: Open-Label Phase Part 1
Description: Adapted JIA ACR 30,50,70,90,100 response=absence of fever due to sJIA in preceding 7 days along with improvement of >=30,50,70,90,100%, respectively in at least 3 out of 6 JIA core set variables with no more than 1 JIA core set variable worsening by >=30%.Variables included: number of joints with active arthritis(any joint with swelling, or absence of swelling, limitation of motion accompanied by either pain on motion or tenderness);number of joints with limited range of motion; physician global evaluation of disease activity on VAS from 0=no disease activity to 10=very severe disease activity, higher scores: greater disease activity; parent/legal guardian/child evaluation of overall well-being on VAS from 0=very well to 10mm=very poor, higher scores: worsen condition; functional ability (Disability Index ranged from 0=no or minimal physical dysfunction, 3=very severe physical dysfunction, higher scores: more physical dysfunction; ESR (mm/hr).
Time Frame: Part 1 Day 7, Part 1 Weeks 2, 4, 8, 12, and 16
Population: OLPT1 analysis set included all participants enrolled into the OL part 1 phase and received at least 1 dose of investigational product in part 1. All participants reported as 'Number of participants analyzed' contributed data to table; but may not have evaluable data for every row. Here, "Number analyzed" participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tofacitinib 5mg BID OL Part 1: Participants were administered tofacitinib 5 mg BID via the oral route and continued to receive a stable dose of Cs during open label part 1.
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of participants
  ACR30: Part 1 Day 7: number analyzed (Participants) | 99
  ACR30: Part 1 Day 7 | 26.26 [17.59 to 34.93]
  ACR30: Part 1 Week 2: number analyzed (Participants) | 99
  ACR30: Part 1 Week 2 | 42.42 [32.69 to 52.16]
  ACR30: Part 1 Week 4: number analyzed (Participants) | 97
  ACR30: Part 1 Week 4 | 68.04 [58.76 to 77.32]
  ACR30: Part 1 Week 8: number analyzed (Participants) | 82
  ACR30: Part 1 Week 8 | 86.59 [79.21 to 93.96]
  ACR30:Part 1 Week 12: number analyzed (Participants) | 44
  ACR30:Part 1 Week 12 | 90.91 [82.41 to 99.40]
  ACR30: Part 1 Week 16: number analyzed (Participants) | 24
  ACR30: Part 1 Week 16 | 83.33 [68.42 to 98.24]
  ACR50:Part 1 Day 7: number analyzed (Participants) | 99
  ACR50:Part 1 Day 7 | 18.18 [10.58 to 25.78]
  ACR50:Part 1 Week 2: number analyzed (Participants) | 99
  ACR50:Part 1 Week 2 | 28.28 [19.41 to 37.15]
  ACR50:Part 1 Week 4: number analyzed (Participants) | 97
  ACR50:Part 1 Week 4 | 44.33 [34.44 to 54.22]
  ACR50:Part 1 Week 8: number analyzed (Participants) | 83
  ACR50:Part 1 Week 8 | 59.04 [48.46 to 69.62]
  ACR50:Part 1 Week 12: number analyzed (Participants) | 44
  ACR50:Part 1 Week 12 | 79.55 [67.63 to 91.46]
  ACR50:Part 1 Week 16: number analyzed (Participants) | 24
  ACR50:Part 1 Week 16 | 75.00 [57.68 to 92.32]
  ACR70:Part 1 Day 7: number analyzed (Participants) | 99
  ACR70:Part 1 Day 7 | 10.10 [4.16 to 16.04]
  ACR70:Part 1 Week 2: number analyzed (Participants) | 99
  ACR70:Part 1 Week 2 | 16.16 [8.91 to 23.41]
  ACR70:Part 1 Week 4: number analyzed (Participants) | 97
  ACR70:Part 1 Week 4 | 19.59 [11.69 to 27.49]
  ACR70:Part 1 Week 8: number analyzed (Participants) | 82
  ACR70:Part 1 Week 8 | 34.15 [23.88 to 44.41]
  ACR70:Part 1 Week 12: number analyzed (Participants) | 44
  ACR70:Part 1 Week 12 | 38.64 [24.25 to 53.02]
  ACR70:Part 1 Week 16: number analyzed (Participants) | 24
  ACR70:Part 1 Week 16 | 33.33 [14.47 to 52.19]
  ACR90:Part 1 Day 7: number analyzed (Participants) | 99
  ACR90:Part 1 Day 7 | 5.05 [0.74 to 9.36]
  ACR90:Part 1 Week 2: number analyzed (Participants) | 99
  ACR90:Part 1 Week 2 | 6.06 [1.36 to 10.76]
  ACR90:Part 1 Week 4: number analyzed (Participants) | 97
  ACR90:Part 1 Week 4 | 11.34 [5.03 to 17.65]
  ACR90:Part 1 Week 8: number analyzed (Participants) | 82
  ACR90:Part 1 Week 8 | 18.29 [9.92 to 26.66]
  ACR90:Part 1 Week 12: number analyzed (Participants) | 44
  ACR90:Part 1 Week 12 | 15.91 [5.10 to 26.72]
  ACR90:Part 1 Week 16: number analyzed (Participants) | 24
  ACR90:Part 1 Week 16 | 16.67 [1.76 to 31.58]
  ACR100:Part 1 Day 7: number analyzed (Participants) | 99
  ACR100:Part 1 Day 7 | 3.03 [0 to 6.41]
  ACR100:Part 1 Week 2: number analyzed (Participants) | 99
  ACR100:Part 1 Week 2 | 5.05 [0.74 to 9.36]
  ACR100:Part 1 Week 4: number analyzed (Participants) | 97
  ACR100:Part 1 Week 4 | 8.25 [2.77 to 13.72]
  ACR100:Part 1 Week 8: number analyzed (Participants) | 82
  ACR100:Part 1 Week 8 | 13.41 [6.04 to 20.79]
  ACR100:Part 1 Week 12: number analyzed (Participants) | 44
  ACR100:Part 1 Week 12 | 9.09 [0.60 to 17.59]
  ACR100:Part 1 Week 16: number analyzed (Participants) | 24
  ACR100:Part 1 Week 16 | 8.33 [0 to 19.39]

7. Secondary Outcome: Percentage of Participants With Adapted JIA ACR 30/50/70/90/100 Response at Part 2 Weeks 4, 8, 12, 16, 20 and 24: Open-label Phase Part 2
Description: as for outcome 6
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20 and 24
Population: OLPT2 analysis set included all participants enrolled into the OL part 2 phase and received at least 1 dose of investigational product in part 1. All participants reported as 'Number of participants analyzed' contributed data to table; but may not have evaluable data for every row. Here, "Number analyzed": participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants
  ACR30:Part 2 Week 4: number analyzed (Participants) | 50
  ACR30:Part 2 Week 4 | 90.00 [81.68 to 98.32]
  ACR30:Part 2 Week 8: number analyzed (Participants) | 40
  ACR30:Part 2 Week 8 | 87.50 [77.25 to 97.75]
  ACR30:Part 2 Week 12: number analyzed (Participants) | 31
  ACR30:Part 2 Week 12 | 90.32 [79.91 to 100]
  ACR30:Part 2 week 16: number analyzed (Participants) | 23
  ACR30:Part 2 week 16 | 86.96 [73.19 to 100]
  ACR30:Part 2 Week 20: number analyzed (Participants) | 13
  ACR30:Part 2 Week 20 | 100 [100 to 100]
  ACR30:Part 2 Week 24: number analyzed (Participants) | 3
  ACR30:Part 2 Week 24 | 100 [100 to 100]
  ACR50:Part 2 Week 4: number analyzed (Participants) | 50
  ACR50:Part 2 Week 4 | 86.00 [76.38 to 95.62]
  ACR50:Part 2 Week 8: number analyzed (Participants) | 40
  ACR50:Part 2 Week 8 | 77.50 [64.56 to 90.44]
  ACR50:Part 2 Week 12: number analyzed (Participants) | 31
  ACR50:Part 2 Week 12 | 80.65 [66.74 to 94.55]
  ACR50:Part 2 Week 16: number analyzed (Participants) | 23
  ACR50:Part 2 Week 16 | 73.91 [55.97 to 91.86]
  ACR50:Part 2 Week 20: number analyzed (Participants) | 13
  ACR50:Part 2 Week 20 | 92.31 [77.82 to 100]
  ACR50:Part 2 Week 24: number analyzed (Participants) | 3
  ACR50:Part 2 Week 24 | 100 [100 to 100]
  ACR70:Part 2 Week 4: number analyzed (Participants) | 50
  ACR70:Part 2 Week 4 | 68.00 [55.07 to 80.93]
  ACR70:Part 2 Week 8: number analyzed (Participants) | 40
  ACR70:Part 2 Week 8 | 67.50 [52.98 to 82.02]
  ACR70:Part 2 Week 12: number analyzed (Participants) | 31
  ACR70:Part 2 Week 12 | 70.97 [54.99 to 86.95]
  ACR70:Part 2 Week 16: number analyzed (Participants) | 23
  ACR70:Part 2 Week 16 | 73.91 [55.97 to 91.86]
  ACR70:Part 2 Week 20: number analyzed (Participants) | 13
  ACR70:Part 2 Week 20 | 92.31 [77.82 to 100]
  ACR70:Part 2 Week 24: number analyzed (Participants) | 3
  ACR70:Part 2 Week 24 | 66.67 [13.32 to 100]
  ACR90:Part 2 Week 4: number analyzed (Participants) | 50
  ACR90:Part 2 Week 4 | 32.00 [19.07 to 44.93]
  ACR90:Part 2 Week 8: number analyzed (Participants) | 40
  ACR90:Part 2 Week 8 | 27.50 [13.66 to 41.34]
  ACR90:Part 2 Week 12: number analyzed (Participants) | 31
  ACR90:Part 2 Week 12 | 22.58 [7.86 to 37.30]
  ACR90:Part 2 Week 16: number analyzed (Participants) | 23
  ACR90:Part 2 Week 16 | 34.78 [15.32 to 54.25]
  ACR90:Part 2 Week 20: number analyzed (Participants) | 13
  ACR90:Part 2 Week 20 | 53.85 [26.75 to 80.95]
  ACR90:Part 2 Week 24: number analyzed (Participants) | 3
  ACR90:Part 2 Week 24 | 33.33 [0 to 86.68]
  ACR100:Part 2 Week 4: number analyzed (Participants) | 50
  ACR100:Part 2 Week 4 | 28.00 [15.55 to 40.45]
  ACR100:Part 2 Week 8: number analyzed (Participants) | 40
  ACR100:Part 2 Week 8 | 27.50 [13.66 to 41.34]
  ACR100:Part 2 Week 12: number analyzed (Participants) | 31
  ACR100:Part 2 Week 12 | 16.13 [3.18 to 29.08]
  ACR100:Part 2 Week 16: number analyzed (Participants) | 23
  ACR100:Part 2 Week 16 | 26.09 [8.14 to 44.03]
  ACR100:Part 2 Week 20: number analyzed (Participants) | 13
  ACR100:Part 2 Week 20 | 38.46 [12.01 to 64.91]
  ACR100:Part 2 Week 24: number analyzed (Participants) | 3
  ACR100:Part 2 Week 24 | 33.33 [0 to 86.68]

8. Secondary Outcome: Percentage of Participants With Fever Attributed to sJIA at Part 1 Days 3, 7 and 14: Open-Label Phase Part 1
Description: Fever was defined as an oral temperature of ˃38 degree Celsius/100.4 degree Fahrenheit. 95% CI was based on normal approximation.
Time Frame: Part 1 Days 3, 7 and 14
Population: OLPT1 analysis set included all participants who were enrolled into the OL part 1 phase of the study and received at least one dose of investigational product in part 1. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies participants evaluable for the specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tofacitinib 5mg BID OL Part 1: Participants were administered tofacitinib 5 mg BID via the oral route and continued to receive a stable dose of Cs during OL part 1.
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of participants
  Part 1 Day 3: number analyzed (Participants) | 96
  Part 1 Day 3 | 3.13 [0 to 6.61]
  Part 1 Day 7: number analyzed (Participants) | 97
  Part 1 Day 7 | 1.03 [0 to 3.04]
  Part 1 Day 14: number analyzed (Participants) | 97
  Part 1 Day 14 | 4.12 [0.17 to 8.08]

9. Secondary Outcome: Percentage of Participants With C-Reactive Protein (CRP) <= 10 mg/L at Baseline, Part 1 Days 3, 7, Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: Percentage of participants with CRP <= 10 milligrams per liter (mg/L) along with 95% CI based on normal approximation is reported in this outcome.
Time Frame: Baseline (last value collected prior to Day 1 of study treatment), Part 1 Days 3, 7, Part 1 Weeks 2, 4, 8, 12, 16
Population: OLPT1 analysis set included all participants who were enrolled into the OL part 1 phase of the study and received at least one dose of investigational product in part 1. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies participants evaluable for the specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of participants
  Baseline | 30.00 [21.02 to 38.98]
  Part 1 Day 3: number analyzed (Participants) | 95
  Part 1 Day 3 | 32.63 [23.20 to 42.06]
  Part 1 Day 7: number analyzed (Participants) | 97
  Part 1 Day 7 | 45.36 [35.45 to 55.27]
  Part 1 Week 2: number analyzed (Participants) | 97
  Part 1 Week 2 | 49.48 [39.53 to 59.43]
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | 55.67 [45.78 to 65.56]
  Part 1 Week 8: number analyzed (Participants) | 80
  Part 1 Week 8 | 60.00 [49.26 to 70.74]
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | 59.09 [44.56 to 73.62]
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | 41.67 [21.94 to 61.39]

10. Secondary Outcome: Percentage of Participants With C-Reactive Protein (CRP) <= 10 mg/L at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-label Phase Part 2
Description: Percentage of participants with CRP <= 10 mg/L along with 95% CI based on normal approximation is reported in this outcome.
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | 68.00 [55.07 to 80.93]
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | 62.50 [47.50 to 77.50]
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | 51.61 [34.02 to 69.21]
  Part 2 Week 16: number analyzed (Participants) | 22
  Part 2 Week 16 | 54.55 [33.74 to 75.35]
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | 76.92 [54.02 to 99.83]
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | 33.33 [0 to 86.68]

11. Secondary Outcome: Percentage of Participants With Absence of Fever Due to sJIA at Part 1 Day 7, Weeks 2, 4, 8, 12, 16: Open-label Phase Part 1
Description: Percentage of participants with absence of fever along with 95% CI based on normal approximation is reported in this outcome.
Time Frame: Part 1 Day 7, Part 1 Weeks 2, 4, 8, 12, 16
Population: OLPT1 analysis set included all participants who were enrolled into the OL part 1 phase of the study and received at least one dose of investigational product in part 1. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of participants
  Part 1 Day 7: number analyzed (Participants) | 97
  Part 1 Day 7 | 83.51 [76.12 to 90.89]
  Part 1 Week 2: number analyzed (Participants) | 97
  Part 1 Week 2 | 82.47 [74.91 to 90.04]
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | 90.72 [84.95 to 96.50]
  Part 1 Week 8: number analyzed (Participants) | 83
  Part 1 Week 8 | 96.39 [92.37 to 100]
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | 100 [100 to 100]
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | 95.83 [87.84 to 100]

12. Secondary Outcome: Percentage of Participants With Absence of Fever Due to sJIA at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 11
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20 and 24
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | 98.00 [94.12 to 100]
  Part 2 Week 8: number analyzed (Participants) | 39
  Part 2 Week 8 | 92.31 [83.94 to 100]
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | 96.77 [90.55 to 100]
  Part 2 Week 16: number analyzed (Participants) | 22
  Part 2 Week 16 | 90.91 [78.90 to 100]
  Part 2 Week 20: number analyzed (Participants) | 12
  Part 2 Week 20 | 100 [100 to 100]
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | 100 [100 to 100]

13. Secondary Outcome: Percentage of Participants With Absence of Fever Due to sJIA at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52: Double Blind Phase
Description: Percentage of participants with absence of fever due sJIA is reported in this outcome. Missing response was imputed as non-response.
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage of participants
  DB Week 4 | 85.71 [72.75 to 98.68] | 93.55 [84.90 to 100]
  DB Week 8 | 85.71 [72.75 to 98.68] | 80.65 [66.74 to 94.55]
  DB Week 12 | 75.00 [58.96 to 91.04] | 74.19 [58.79 to 89.60]
  DB Week 16 | 71.43 [54.70 to 88.16] | 61.29 [44.14 to 78.44]
  DB Week 20 | 67.86 [50.56 to 85.16] | 51.61 [34.02 to 69.21]
  DB Week 24 | 64.29 [46.54 to 82.03] | 54.84 [37.32 to 72.36]
  DB Week 28 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  DB Week 32 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  DB Week 36 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  DB Week 40 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  DB Week 44 | 60.71 [42.62 to 78.80] | 51.61 [34.02 to 69.21]
  DB Week 48 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
  DB Week 52 | 60.71 [42.62 to 78.80] | 48.39 [30.79 to 65.98]
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4; Test type: Other; Difference in percentage = -7.83, 95% CI 2-sided [-23.42 to 7.75] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8; Test type: Other; Difference in percentage = 5.07, 95% CI 2-sided [-13.94 to 24.08] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12; Test type: Other; Difference in percentage = 0.81, 95% CI 2-sided [-21.43 to 23.04] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16; Test type: Other; Difference in percentage = 10.14, 95% CI 2-sided [-13.82 to 34.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20; Test type: Other; Difference in percentage = 16.24, 95% CI 2-sided [-8.43 to 40.92] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24; Test type: Other; Difference in percentage = 9.45, 95% CI 2-sided [-15.49 to 34.39] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44; Test type: Other; Difference in percentage = 9.10, 95% CI 2-sided [-16.13 to 34.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52; Test type: Other; Difference in percentage = 12.33, 95% CI 2-sided [-12.91 to 37.56] — [estimate comment as in outcome 5, analysis 1]

14. Secondary Outcome: Time to First Adapted JIA ACR 30 Response: Open-label Phase Part 1
Description: Time to the first adapted JIA ACR 30 response was measured in number of days since Day 1 (day of adapted JIA ACR 30 response - Day 1 + 1) in the OL Phase Part 1. Participants that did not achieve an adapted JIA ACR30 response defined as absence of fever due to sJIA [temperature =<38 degree Celsius/100.4 degree F in the preceding 7 days along with an improvement of at least 30% from baseline (Day 1 of study drug before first tofacitinib administration) in at least 3 of the 6 JIA core components, with worsening of >=30 in no more than 1 of the remaining components, which in Part 1 (withdrew from the study) were censored at their last available response assessment in Part 1. 95% CI was based on the Brookmeyer and Crowley Method.
Time Frame: From Day 1 up to 16 weeks
Population: OLPT1 analysis set included all participants who were enrolled into the OP part 1 phase of the study and received at least one dose of investigational product in part 1.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Days | 27.0 [15.0 to 29.0]

15. Secondary Outcome: Change From Open Label Baseline in Juvenile Arthritis Disease Activity Score (JADAS-27) Erythrocyte Sedimentation Rate (ESR) at Part 1 Day 7, Part 1 Weeks 2, 4, 8, 12 and 16: Open-Label Phase Part 1
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 ESR score was determined based on four components: Physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ) assessed on a VAS of 0 [very well] to 10 [very poor], ESR (value normalized to 0 to 10 scale) and number of joints with active disease (27 joint assessment ranging from 0 to 27). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57. A higher score indicated more disease activity.
Time Frame: Baseline (last value collected prior to day 1 of tofacitinib administration in OL phase), Part 1 Day 7, Part 1 Weeks 2, 4, 8, 12 and 16
Population: OLPT1 analysis set included all participants who were enrolled into the OL part 1 phase of the study and received at least one dose of investigational product in part 1. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Units on a scale
  Part 1 Day 7: number analyzed (Participants) | 98
  Part 1 Day 7 | -5.64 (5.20)
  Part 1 Week 2: number analyzed (Participants) | 98
  Part 1 Week 2 | -8.57 (5.97)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -11.95 (6.53)
  Part 1 Week 8: number analyzed (Participants) | 81
  Part 1 Week 8 | -15.09 (7.27)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -15.77 (7.24)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -14.08 (6.09)

16. Secondary Outcome: Change From Open-Label Baseline in JADAS-27 CRP at Part 1 Day 7, Part 1 Weeks 2, 4, 8, 12 and 16: Open-Label Phase Part 1
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 CRP score was determined based on four components: physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 [very well] to 10 [very poor]), CRP (value normalized to 0 to 10 scale) and number of joints with active disease (27 joint assessment ranging from 0 to 27). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57. A higher score indicated more disease activity.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Units on a scale
  Part 1 Day 7: number analyzed (Participants) | 97
  Part 1 Day 7 | -6.25 (5.53)
  Part 1 Week 2: number analyzed (Participants) | 96
  Part 1 Week 2 | -8.55 (6.10)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -11.88 (7.28)
  Part 1 Week 8: number analyzed (Participants) | 80
  Part 1 Week 8 | -15.07 (8.46)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -15.19 (7.73)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -13.10 (6.37)

17. Secondary Outcome: Change From Open-Label Baseline in JADAS-27 ESR at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 ESR score was determined based on four components: physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 [very well] to 10 [very poor]), ESR (value normalized to 0 to 10 scale) and number of joints with active disease (27 joint assessment ranging from 0 to 27). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57. A higher score indicated more disease activity.
Time Frame: Baseline (last value collected prior to day 1 of tofacitinib administration in OL phase), Part 2 Weeks 4, 8, 12, 16, 20 and 24
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Units on a scale
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -17.05 (8.18)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -17.13 (8.14)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -18.17 (7.74)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -18.89 (7.56)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -21.14 (5.78)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -22.17 (7.58)

18. Secondary Outcome: Change From Open-Label Baseline in JADAS-27 CRP at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 16
Time Frame: as for outcome 17
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Units on a scale
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -17.16 (8.87)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -17.44 (8.03)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -18.99 (7.67)
  Part 2 Week 16: number analyzed (Participants) | 22
  Part 2 Week 16 | -20.31 (6.41)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -22.16 (7.05)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -25.61 (9.82)

19. Secondary Outcome: Change From Double-Blind Baseline in JADAS-27 ESR at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 ESR score was determined based on four components: Physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ) (assessed on a VAS of 0 [very well] to 10 [very poor]), ESR (value normalized to 0 to 10 scale) and number of joints with active disease (27 joint assessment ranging from 0 to 27). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57. A higher score indicated more disease activity.
Time Frame: DB Baseline (at randomization on Day 1 in DB phase), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: DBFAS consisted of all randomized participants who received at least one dose of investigational product in the DB phase. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 30
  DB Week 4 | 1.07 (0.84) | 1.08 (0.79)
  DB Week 8: number analyzed (Participants) | 25 | 24
  DB Week 8 | 1.75 (1.08) | 0.81 (1.06)
  DB Week 12: number analyzed (Participants) | 21 | 22
  DB Week 12 | 1.47 (1.46) | 1.71 (1.40)
  DB Week 16: number analyzed (Participants) | 21 | 19
  DB Week 16 | 0.43 (1.03) | 1.29 (1.04)
  DB Week 20: number analyzed (Participants) | 19 | 14
  DB Week 20 | -1.04 (0.65) | 0.05 (0.69)
  DB Week 24: number analyzed (Participants) | 18 | 14
  DB Week 24 | -0.49 (0.57) | -0.79 (0.60)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | 2.58 (2.05) | 3.86 (2.25)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -0.21 (0.77) | -0.68 (0.83)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -1.52 (0.50) | -1.26 (0.54)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -0.23 (0.91) | -0.96 (0.96)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -1.67 (0.75) | -0.83 (0.79)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -2.29 (0.38) | -2.06 (0.60)
  DB Week 52: number analyzed (Participants) | 6 | 4
  DB Week 52 | -2.41 (0.60) | -1.65 (1.07)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.01, 95% CI 2-sided [-2.40 to 2.38]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.94, 95% CI 2-sided [-2.25 to 4.12]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.24, 95% CI 2-sided [-4.54 to 4.06]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.86, 95% CI 2-sided [-3.99 to 2.28]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -1.09, 95% CI 2-sided [-3.12 to 0.94]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.30, 95% CI 2-sided [-1.46 to 2.06]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -1.28, 95% CI 2-sided [-7.85 to 5.29]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.48, 95% CI 2-sided [-1.98 to 2.93]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.26, 95% CI 2-sided [-1.86 to 1.35]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.73, 95% CI 2-sided [-2.18 to 3.63]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.83, 95% CI 2-sided [-3.22 to 1.56]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.23, 95% CI 2-sided [-1.76 to 1.30]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.75, 95% CI 2-sided [-3.43 to 1.93]

20. Secondary Outcome: Change From Double-Blind Baseline in JADAS-27 CRP at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 16
Time Frame: DB Baseline (at randomization on Day 1 in DB phase), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 26 | 31
  DB Week 4 | 1.62 (0.96) | 0.71 (0.90)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | 2.12 (0.95) | 0.01 (0.93)
  DB Week 12: number analyzed (Participants) | 21 | 22
  DB Week 12 | 1.78 (1.46) | 1.80 (1.40)
  DB Week 16: number analyzed (Participants) | 21 | 19
  DB Week 16 | 0.84 (1.09) | 1.95 (1.08)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -0.17 (0.84) | 0.36 (0.87)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | 1.58 (1.04) | -0.26 (1.08)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | 2.64 (1.86) | 2.72 (2.04)
  DB Week 32: number analyzed (Participants) | 12 | 9
  DB Week 32 | 0.49 (0.99) | 1.18 (1.07)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -1.59 (0.50) | -1.24 (0.53)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | 0.38 (1.15) | 0.41 (1.21)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -1.09 (0.99) | 1.50 (1.02)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -2.04 (0.51) | -1.23 (0.76)
  DB Week 52: number analyzed (Participants) | 6 | 4
  DB Week 52 | -2.31 (0.60) | -1.85 (1.10)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 1]; Test type: Other; Difference in LS Mean = 0.90, 95% CI 2-sided [-1.80 to 3.61]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 2]; Test type: Other; Difference in LS Mean = 2.11, 95% CI 2-sided [-0.64 to 4.86]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 3]; Test type: Other; Difference in LS Mean = -0.02, 95% CI 2-sided [-4.25 to 4.21]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 4]; Test type: Other; Difference in LS Mean = -1.12, 95% CI 2-sided [-4.32 to 2.09]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 5]; Test type: Other; Difference in LS Mean = -0.53, 95% CI 2-sided [-3.04 to 1.98]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 6]; Test type: Other; Difference in LS Mean = 1.84, 95% CI 2-sided [-1.29 to 4.97]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 7]; Test type: Other; Difference in LS Mean = -0.08, 95% CI 2-sided [-5.89 to 5.72]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 8]; Test type: Other; Difference in LS Mean = -0.69, 95% CI 2-sided [-3.79 to 2.41]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 9]; Test type: Other; Difference in LS Mean = -0.35, 95% CI 2-sided [-1.89 to 1.19]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 10]; Test type: Other; Difference in LS Mean = -0.03, 95% CI 2-sided [-3.63 to 3.58]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 11]; Test type: Other; Difference in LS Mean = -2.59, 95% CI 2-sided [-5.67 to 0.49]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 12]; Test type: Other; Difference in LS Mean = -0.82, 95% CI 2-sided [-2.82 to 1.19]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 13]; Test type: Other; Difference in LS Mean = -0.46, 95% CI 2-sided [-3.27 to 2.36]

21. Secondary Outcome: Change From Open-Label Baseline in Number of Joints With Active Arthritis at Part 1 Day 7, Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: The ACR defined a joint with active arthritis as a joint with swelling or, in the absence of swelling, limitation of motion accompanied by pain on motion, or tenderness.
Time Frame: as for outcome 15
Population: OLPT1 analysis set included all participants who were enrolled into the OL part 1 phase of the study and received at least one dose of investigational product in part 1. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Joints
  Part 1 Day 7: number analyzed (Participants) | 99
  Part 1 Day 7 | -2.96 (4.17)
  Part 1 Week 2: number analyzed (Participants) | 99
  Part 1 Week 2 | -4.21 (5.31)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -6.03 (6.04)
  Part 1 Week 8: number analyzed (Participants) | 83
  Part 1 Week 8 | -7.80 (9.25)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -7.52 (7.38)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -6.38 (7.87)

22. Secondary Outcome: Change From Open-Label Baseline in Number of Joints With Active Arthritis at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 21
Time Frame: Baseline (last value collected prior to day 1 of tofacitinib administration in OL phase), Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Joints
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -7.78 (7.78)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -7.73 (8.40)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -9.26 (7.98)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -10.00 (7.99)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -10.85 (7.83)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -13.67 (11.02)

23. Secondary Outcome: Change From Open-Label Baseline in Number of Joints With Limited Range of Motion at Part 1 Day 7, Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: Limitation of motion were assessed in the following joints: Temporomandibular, shoulder, elbow, wrist, metacarpophalangeal (MCP I-V), proximal interphalangeal (PIP I-V), distal interphalangeal (II-V), hip, knee, ankle, subtalar joints, intertarsal joints, metatarsophalangeal (MTP I-V), toe interphalangeal (I-V), cervical spine, thoracic spine, lumbar spine.
Time Frame: Baseline (last value collected prior to day 1 of tofacitinib administration in OL phase), Part 1 Day 7, Weeks 2, 4, 8, 12, 16
Population: OLPT1 analysis set included all participants who were enrolled into the OL part 1 phase of the study and received at least one dose of investigational product in part 1. All participants reported under 'Number of participants analyzed contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Joints
  Part 1 Day 7: number analyzed (Participants) | 99
  Part 1 Day 7 | -1.83 (4.26)
  Part 1 Week 2: number analyzed (Participants) | 99
  Part 1 Week 2 | -2.06 (4.70)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -2.90 (5.42)
  Part 1 Week 8: number analyzed (Participants) | 83
  Part 1 Week 8 | -4.36 (8.59)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -3.64 (6.05)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -2.33 (3.48)

24. Secondary Outcome: Change From Open-Label Baseline in Number of Joints With Limited Range of Motion at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 23
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Joints
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -4.26 (6.75)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -3.90 (6.08)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -5.81 (7.48)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -5.74 (7.13)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -5.92 (9.32)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -15.67 (11.02)

25. Secondary Outcome: Change From Open-Label Baseline in Physician Global Evaluation of Disease Activity at Part 1 Day 7, Weeks 2, 4, 8, 12, 16: Open-label Phase Part 1
Description: Physician global evaluation of disease activity was assessed on a 21-numbered circle VAS ranging from 0 to 10, where 0= no disease activity and 10= maximum disease activity. Where higher scores indicated more disease activity.
Time Frame: as for outcome 23
Population: OLPT1 analysis set included all participants who were enrolled into the OL part 1 phase of the study and received at least one dose of investigational product in part 1. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
units on a scale
  Part 1 Day 7: number analyzed (Participants) | 99
  Part 1 Day 7 | -1.18 (1.36)
  Part 1 Week 2: number analyzed (Participants) | 99
  Part 1 Week 2 | -1.82 (1.68)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -2.62 (1.75)
  Part 1 Week 8: number analyzed (Participants) | 83
  Part 1 Week 8 | -3.40 (2.01)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -3.66 (2.08)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -3.50 (1.93)

26. Secondary Outcome: Change From Open-Label Baseline in Physician Global Evaluation of Disease Activity at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 25
Time Frame: as for outcome 22
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Unit on a scale
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -4.54 (2.10)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -4.53 (1.74)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -4.65 (1.57)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -4.89 (1.77)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -5.62 (1.21)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -6.17 (1.44)

27. Secondary Outcome: Change From Open-Label Baseline in ESR at Part 1 Day 7, Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: ESR was determined using an ESR testing kit.
Time Frame: as for outcome 23
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Millimeter per hour
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Millimeter per hour
  Part 1 Day 7: number analyzed (Participants) | 98
  Part 1 Day 7 | -11.00 (16.96)
  Part 1 Week 2: number analyzed (Participants) | 99
  Part 1 Week 2 | -18.60 (19.78)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -24.70 (23.86)
  Part 1 Week 8: number analyzed (Participants) | 81
  Part 1 Week 8 | -30.59 (23.12)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -31.74 (21.75)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -27.65 (28.84)

28. Secondary Outcome: Change From Open-Label Baseline in ESR at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: ESR was determined using an ESR testing kit.
Time Frame: as for outcome 22
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimeter per hour
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Millimeter per hour
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -33.64 (28.16)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -30.73 (27.11)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -27.52 (28.13)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -23.48 (24.70)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -37.54 (20.93)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -24.33 (6.03)

29. Secondary Outcome: Change From Open-Label Baseline in CHAQ- Parental Evaluation of Overall Well-being at Part 1 Days 3, 7, Part 1 Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: The CHAQ, derived from the adult health assessment questionnaire, comprised of two indices disability and discomfort, and parent global assessment of overall well-being. For assessment of overall well-being, the parent/legal guardian/participant were required to rate the overall well-being by entering a number from 0 to 10 (in 0.5 increments), on a 21-circle VAS where '0= very well and 10=very poorly. Where higher scores indicated worse condition.
Time Frame: Baseline (last value collected prior to day 1 of tofacitinib administration in OL phase), Part 1 Days 3,7, Part 1 Weeks 2, 4, 8, 12, 16
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Units on a scale
  Part 1 Day 3: number analyzed (Participants) | 96
  Part 1 Day 3 | -0.73 (1.53)
  Part 1 Day 7: number analyzed (Participants) | 99
  Part 1 Day 7 | -1.36 (1.91)
  Part 1 Week 2: number analyzed (Participants) | 98
  Part 1 Week 2 | -1.96 (1.89)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -2.65 (2.44)
  Part 1 Week 8: number analyzed (Participants) | 83
  Part 1 Week 8 | -3.35 (2.38)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -3.45 (2.45)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -3.48 (2.78)

30. Secondary Outcome: Change From Open-Label Baseline in CHAQ - Parental Evaluation of Overall Well-being at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: The CHAQ, derived from the adult health assessment questionnaire, comprised of two indices disability and discomfort, and parent global assessment of overall well-being. For assessment of overall well-being, the parent/legal guardian/participant were required to rate the overall well-being by entering a number from 0 to 10 (in 0.5 increments), on a 21-circle VAS where '0=Very Well and 10=Very Poorly. Where higher scores indicated worse condition.
Time Frame: as for outcome 22
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Units on a scale
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -4.09 (2.68)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -4.50 (2.88)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -4.73 (2.83)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -5.11 (2.50)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -5.65 (2.89)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -6.33 (2.31)

31. Secondary Outcome: Change From Open-Label Baseline in CHAQ - Disability Index at Part 1 Day 7, Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: CHAQ, derived from the adult health assessment questionnaire, comprised of two indices disability and discomfort, and parent global assessment of overall Well-being. CHAQ disability index consisted of 30 items in 8 areas: 1. dressing and grooming, 2. arising, 3. eating, 4. walking, 5. hygiene, 6. reach, 7. grip, and 8. activities distributed. Each item was rated on a 4-point scale, scored from 0 (no difficulty) to 3 (unable to do). The eight areas of the CHAQ were averaged to calculate the total disability index score which ranged from 0 (no or minimal physical dysfunction) to 3 (very severe physical dysfunction), higher scores indicated more disability. A participant must have score for at least six of the eight areas, otherwise a CHAQ-DI score was not valid.
Time Frame: as for outcome 23
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Units on a scale
  Part 1 Day 7: number analyzed (Participants) | 99
  Part 1 Day 7 | -0.21 (0.35)
  Part 1 Week 2: number analyzed (Participants) | 99
  Part 1 Week 2 | -0.38 (0.43)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -0.52 (0.56)
  Part 1 Week 8: number analyzed (Participants) | 83
  Part 1 Week 8 | -0.59 (0.57)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -0.51 (0.56)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -0.74 (0.73)

32. Secondary Outcome: Change From Open-Label Baseline in CHAQ-Disability Index at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: CHAQ, derived from the adult health assessment questionnaire, comprised of two indices disability and discomfort, and parent global assessment of overall well-being. CHAQ disability index consisted of 30 items in 8 areas, 1. dressing and grooming, 2. arising, 3. eating, 4. walking, 5. hygiene, 6. reach, 7. grip, and 8. activities distributed. Each item was rated on a 4-point scale, scored from 0 (no difficulty) to-3 (unable to do). The eight areas of the CHAQ were averaged to calculate the total disability index score which ranged from 0 (no or minimal physical dysfunction) to 3 (very severe physical dysfunction), higher scores indicated more disability. A participant must have score for at least six of the eight areas, otherwise a CHAQ-DI score was not valid.
Time Frame: as for outcome 22
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 1. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Units on a scale
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -0.79 (0.63)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -0.78 (0.76)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -0.85 (0.80)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -0.67 (0.74)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -0.93 (0.77)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -0.96 (0.92)

33. Secondary Outcome: Change From Open-Label Baseline in Number of Joints With Active Arthritis at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 21
Time Frame: OL Baseline (last value collected prior to Day 1 of tofacitinib administration in OL phase), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: DBFAS consisted of all randomized participants who received at least one dose of investigational product in the DB phase. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Joints
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | -6.53 (0.34) | -7.39 (0.32)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | -6.36 (0.38) | -7.69 (0.38)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | -5.92 (0.80) | -7.36 (0.76)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -7.34 (0.25) | -7.37 (0.25)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -7.41 (0.18) | -7.51 (0.20)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -7.33 (0.13) | -7.76 (0.13)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -6.36 (0.59) | -6.56 (0.67)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -7.27 (0.17) | -7.76 (0.19)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -7.43 (0.14) | -7.78 (0.16)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -7.06 (0.24) | -7.58 (0.27)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -7.39 (0.33) | -7.20 (0.35)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -7.54 (0.20) | -7.75 (0.25)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -7.46 (0.26) | -7.51 (0.28)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 4: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.86, 95% CI 2-sided [-0.08 to 1.79]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 8: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 1.32, 95% CI 2-sided [0.25 to 2.40]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 12: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 1.43, 95% CI 2-sided [-0.79 to 3.66]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 16: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.02, 95% CI 2-sided [-0.70 to 0.74]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 20: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.11, 95% CI 2-sided [-0.43 to 0.64]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.44, 95% CI 2-sided [0.06 to 0.81]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 28: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.21, 95% CI 2-sided [-1.64 to 2.06]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 32: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.49, 95% CI 2-sided [-0.04 to 1.03]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 36: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.35, 95% CI 2-sided [-0.09 to 0.79]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 40: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.52, 95% CI 2-sided [-0.23 to 1.28]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 44: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.19, 95% CI 2-sided [-1.20 to 0.83]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.21, 95% CI 2-sided [-0.49 to 0.91]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 52: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open-Label baseline value, and Open-Label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.06, 95% CI 2-sided [-0.80 to 0.92]

34. Secondary Outcome: Change From Double-Blind Baseline in Number of Joints With Active Arthritis at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 21
Time Frame: DB Baseline (randomization), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Joints
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | 0.38 (0.26) | 0.09 (0.24)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | 0.78 (0.38) | -0.23 (0.37)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | 1.47 (0.85) | 0.22 (0.81)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | 0.05 (0.27) | -0.05 (0.27)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -0.15 (0.15) | -0.02 (0.17)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -0.06 (0.12) | -0.39 (0.13)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | 0.71 (0.70) | 0.88 (0.84)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | 0.01 (0.18) | -0.41 (0.20)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -0.14 (0.15) | -0.47 (0.17)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | 0.31 (0.25) | -0.37 (0.28)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -0.05 (0.35) | 0.11 (0.38)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -0.20 (0.21) | -0.56 (0.27)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -0.14 (0.28) | -0.38 (0.34)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 1]; Test type: Other; Difference in LS Mean = 0.29, 95% CI 2-sided [-0.43 to 1.00]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 2]; Test type: Other; Difference in LS Mean = 1.01, 95% CI 2-sided [-0.06 to 2.08]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 3]; Test type: Other; Difference in LS Mean = 1.25, 95% CI 2-sided [-1.13 to 3.64]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 4]; Test type: Other; Difference in LS Mean = 0.10, 95% CI 2-sided [-0.68 to 0.88]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 5]; Test type: Other; Difference in LS Mean = -0.13, 95% CI 2-sided [-0.58 to 0.33]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 6]; Test type: Other; Difference in LS Mean = 0.32, 95% CI 2-sided [-0.03 to 0.68]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 7]; Test type: Other; Difference in LS Mean = -0.17, 95% CI 2-sided [-2.42 to 2.08]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 8]; Test type: Other; Difference in LS Mean = 0.42, 95% CI 2-sided [-0.14 to 0.97]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 9]; Test type: Other; Difference in LS Mean = 0.32, 95% CI 2-sided [-0.15 to 0.79]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 10]; Test type: Other; Difference in LS Mean = 0.68, 95% CI 2-sided [-0.14 to 1.49]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 11]; Test type: Other; Difference in LS Mean = -0.16, 95% CI 2-sided [-1.28 to 0.96]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 12]; Test type: Other; Difference in LS Mean = 0.37, 95% CI 2-sided [-0.43 to 1.16]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 13]; Test type: Other; Difference in LS Mean = 0.24, 95% CI 2-sided [-0.82 to 1.30]

35. Secondary Outcome: Change From Open-Label Baseline in CHAQ-Disability Index at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: The parents were asked to provide responses to questions designed to assessed function in 8 distributed, among a total of 30 items. Each question was rated on a four-point scale, scored from 0-3. The question with the highest score determined the score for the functional area. If aids or devices were used or assistance was required, the minimum score for that was 2. Each question was rated 0 for no difficulty, 1 for some difficulties, 2 for much difficulties, and 3 for unable to do. The 8 areas of the CHAQ were averaged to calculated disability index which was ranges from 0 (no or minimal physical dysfunction) to 3 (very severe physical dysfunction). A participant must have score for at least 6 of the 8 categories, otherwise a CHAQ-DI score was not valid.
Time Frame: as for outcome 33
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | -0.81 (0.10) | -1.03 (0.09)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | -0.93 (0.08) | -1.02 (0.08)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | -0.99 (0.08) | -1.04 (0.07)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -0.95 (0.09) | -1.05 (0.09)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -1.02 (0.07) | -1.21 (0.07)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -0.94 (0.08) | -1.05 (0.08)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -0.94 (0.08) | -1.01 (0.09)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -0.96 (0.07) | -1.11 (0.07)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -1.05 (0.08) | -1.16 (0.09)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -1.07 (0.07) | -1.22 (0.08)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -1.04 (0.09) | -1.08 (0.09)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -1.01 (0.09) | -1.10 (0.11)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -1.04 (0.10) | -1.13 (0.12)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 1]; Test type: Other; Difference in LS Mean = 0.21, 95% CI 2-sided [-0.07 to 0.50]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 2]; Test type: Other; Difference in LS Mean = 0.09, 95% CI 2-sided [-0.15 to 0.32]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 3]; Test type: Other; Difference in LS Mean = 0.05, 95% CI 2-sided [-0.17 to 0.28]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 4]; Test type: Other; Difference in LS Mean = 0.10, 95% CI 2-sided [-0.16 to 0.36]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 5]; Test type: Other; Difference in LS Mean = 0.19, 95% CI 2-sided [-0.01 to 0.38]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 6]; Test type: Other; Difference in LS Mean = 0.12, 95% CI 2-sided [-0.12 to 0.35]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 7]; Test type: Other; Difference in LS Mean = 0.07, 95% CI 2-sided [-0.18 to 0.31]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 8]; Test type: Other; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.06 to 0.37]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 9]; Test type: Other; Difference in LS Mean = 0.11, 95% CI 2-sided [-0.14 to 0.36]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 10]; Test type: Other; Difference in LS Mean = 0.16, 95% CI 2-sided [-0.06 to 0.38]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 11]; Test type: Other; Difference in LS Mean = 0.04, 95% CI 2-sided [-0.22 to 0.30]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 12]; Test type: Other; Difference in LS Mean = 0.09, 95% CI 2-sided [-0.20 to 0.38]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 13]; Test type: Other; Difference in LS Mean = 0.09, 95% CI 2-sided [-0.24 to 0.42]

36. Secondary Outcome: Change From Double Blind Baseline in CHAQ-Disability Index at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 35
Time Frame: DB Baseline (randomization), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: DBFAS consisted of all randomized participants who received at least one dose of investigational product in the DB phase. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | 0.04 (0.06) | -0.02 (0.06)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | -0.03 (0.06) | -0.01 (0.06)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | -0.06 (0.06) | -0.05 (0.06)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -0.03 (0.07) | -0.05 (0.07)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -0.08 (0.06) | -0.23 (0.06)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | 0.06 (0.08) | -0.09 (0.08)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | 0.05 (0.08) | -0.04 (0.09)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | 0.02 (0.07) | -0.13 (0.07)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -0.03 (0.09) | -0.19 (0.09)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -0.09 (0.07) | -0.25 (0.07)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -0.06 (0.09) | -0.10 (0.09)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -0.03 (0.09) | -0.19 (0.12)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -0.05 (0.10) | -0.21 (0.13)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 1]; Test type: Other; Difference in LS Mean = 0.07, 95% CI 2-sided [-0.10 to 0.24]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 2]; Test type: Other; Difference in LS Mean = -0.02, 95% CI 2-sided [-0.19 to 0.15]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 3]; Test type: Other; Difference in LS Mean = -0.01, 95% CI 2-sided [-0.19 to 0.16]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 4]; Test type: Other; Difference in LS Mean = 0.01, 95% CI 2-sided [-0.20 to 0.23]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 5]; Test type: Other; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.02 to 0.32]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 6]; Test type: Other; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.09 to 0.40]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 7]; Test type: Other; Difference in LS Mean = 0.09, 95% CI 2-sided [-0.16 to 0.34]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 8]; Test type: Other; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.05 to 0.36]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 9]; Test type: Other; Difference in LS Mean = 0.16, 95% CI 2-sided [-0.10 to 0.43]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 10]; Test type: Other; Difference in LS Mean = 0.17, 95% CI 2-sided [-0.06 to 0.39]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 11]; Test type: Other; Difference in LS Mean = 0.04, 95% CI 2-sided [-0.22 to 0.30]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 12]; Test type: Other; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.18 to 0.49]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 13]; Test type: Other; Difference in LS Mean = 0.16, 95% CI 2-sided [-0.23 to 0.55]

37. Secondary Outcome: Change From Open-Label Baseline in Number of Joints With Limited Range of Motion at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 23
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Joints
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | -2.47 (0.43) | -2.69 (0.41)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | -2.31 (0.45) | -2.89 (0.44)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | -2.09 (0.71) | -3.29 (0.68)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -2.76 (0.44) | -2.70 (0.43)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -2.79 (0.19) | -3.05 (0.19)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -2.98 (0.19) | -3.07 (0.19)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -2.56 (0.54) | -2.10 (0.56)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -2.89 (0.18) | -3.24 (0.19)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -2.90 (0.19) | -3.21 (0.21)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -2.96 (0.24) | -3.24 (0.25)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -2.95 (0.25) | -3.24 (0.26)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -3.03 (0.27) | -3.25 (0.30)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -2.75 (0.36) | -3.20 (0.36)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 4: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.21, 95% CI 2-sided [-0.97 to 1.40]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 8: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.58, 95% CI 2-sided [-0.68 to 1.84]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 12: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 1.20, 95% CI 2-sided [-0.77 to 3.16]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 16: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.06, 95% CI 2-sided [-1.30 to 1.18]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 20: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.26, 95% CI 2-sided [-0.29 to 0.82]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.09, 95% CI 2-sided [-0.46 to 0.64]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 28: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.46, 95% CI 2-sided [-2.05 to 1.13]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 32: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.35, 95% CI 2-sided [-0.18 to 0.88]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 36: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.31, 95% CI 2-sided [-0.26 to 0.88]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 40: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.28, 95% CI 2-sided [-0.43 to 0.99]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 44: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.29, 95% CI 2-sided [-0.45 to 1.03]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.22, 95% CI 2-sided [-0.63 to 1.08]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB week 52: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Open label baseline value, and Open-label baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.45, 95% CI 2-sided [-0.66 to 1.57]

38. Secondary Outcome: Change From Double-Blind Baseline in Number of Joints With Limited Range of Motion at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 23
Time Frame: DB Baseline (values at randomization), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Joints
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | 0.08 (0.22) | 0.21 (0.20)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | 0.45 (0.42) | 0.06 (0.42)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | 0.48 (0.44) | -0.23 (0.42)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -0.30 (0.17) | 0.10 (0.17)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -0.36 (0.10) | -0.19 (0.11)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -0.53 (0.10) | -0.22 (0.11)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -0.05 (0.40) | 1.05 (0.46)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -0.41 (0.10) | -0.48 (0.12)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -0.48 (0.09) | -0.46 (0.10)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -0.48 (0.15) | -0.43 (0.17)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -0.47 (0.16) | -0.43 (0.17)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -0.50 (0.20) | -0.47 (0.24)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -0.21 (0.31) | -0.42 (0.33)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 1]; Test type: Other; Difference in LS Mean = -0.13, 95% CI 2-sided [-0.73 to 0.47]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 2]; Test type: Other; Difference in LS Mean = 0.39, 95% CI 2-sided [-0.81 to 1.59]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 3]; Test type: Other; Difference in LS Mean = 0.70, 95% CI 2-sided [-0.54 to 1.95]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 4]; Test type: Other; Difference in LS Mean = -0.40, 95% CI 2-sided [-0.90 to 0.10]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 5]; Test type: Other; Difference in LS Mean = -0.16, 95% CI 2-sided [-0.46 to 0.13]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 6]; Test type: Other; Difference in LS Mean = -0.32, 95% CI 2-sided [-0.63 to -0.01]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 7]; Test type: Other; Difference in LS Mean = -1.09, 95% CI 2-sided [-2.34 to 0.15]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 8]; Test type: Other; Difference in LS Mean = 0.07, 95% CI 2-sided [-0.26 to 0.40]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 9]; Test type: Other; Difference in LS Mean = -0.02, 95% CI 2-sided [-0.30 to 0.26]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 10]; Test type: Other; Difference in LS Mean = -0.05, 95% CI 2-sided [-0.53 to 0.43]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 11]; Test type: Other; Difference in LS Mean = -0.05, 95% CI 2-sided [-0.56 to 0.46]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 12]; Test type: Other; Difference in LS Mean = -0.03, 95% CI 2-sided [-0.74 to 0.69]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 13]; Test type: Other; Difference in LS Mean = 0.20, 95% CI 2-sided [-0.91 to 1.32]

39. Secondary Outcome: Change From Open-Label Baseline in Physician Global Evaluation of Disease Activity at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: Physician global evaluation of disease activity was assessed on a 21-numbered circle VAS ranging from 0 to 10, where 0= no disease activity and 10=maximum disease activity, where higher scores indicated more disease activity.
Time Frame: OL label Baseline (last value collected prior to Day 1 of tofacitinib administration in OL phase), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: DBFAS consisted of all randomized participants who received at least one dose of investigational product in the DB phase. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | -4.22 (0.33) | -5.22 (0.32)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | -4.23 (0.32) | -5.55 (0.32)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | -4.89 (0.36) | -5.42 (0.34)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -4.96 (0.32) | -5.22 (0.32)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -5.32 (0.23) | -5.64 (0.24)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -5.11 (0.22) | -5.66 (0.23)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -5.06 (0.37) | -5.26 (0.40)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -5.08 (0.26) | -5.71 (0.28)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -5.55 (0.16) | -6.03 (0.18)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -5.23 (0.30) | -5.88 (0.33)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -5.65 (0.21) | -5.87 (0.22)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -5.87 (0.18) | -6.14 (0.24)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -5.86 (0.26) | -5.97 (0.33)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 1]; Test type: Other; Difference in LS Mean = 1.01, 95% CI 2-sided [0.09 to 1.92]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 2]; Test type: Other; Difference in LS Mean = 1.31, 95% CI 2-sided [0.40 to 2.22]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 3]; Test type: Other; Difference in LS Mean = 0.53, 95% CI 2-sided [-0.47 to 1.53]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 4]; Test type: Other; Difference in LS Mean = 0.26, 95% CI 2-sided [-0.63 to 1.16]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 5]; Test type: Other; Difference in LS Mean = 0.32, 95% CI 2-sided [-0.33 to 0.97]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 6]; Test type: Other; Difference in LS Mean = 0.55, 95% CI 2-sided [-0.10 to 1.20]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 7]; Test type: Other; Difference in LS Mean = 0.20, 95% CI 2-sided [-0.93 to 1.33]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 8]; Test type: Other; Difference in LS Mean = 0.62, 95% CI 2-sided [-0.17 to 1.42]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 9]; Test type: Other; Difference in LS Mean = 0.48, 95% CI 2-sided [-0.02 to 0.98]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 10]; Test type: Other; Difference in LS Mean = 0.64, 95% CI 2-sided [-0.30 to 1.58]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 11]; Test type: Other; Difference in LS Mean = 0.23, 95% CI 2-sided [-0.40 to 0.85]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 12]; Test type: Other; Difference in LS Mean = 0.26, 95% CI 2-sided [-0.36 to 0.88]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 13]; Test type: Other; Difference in LS Mean = 0.11, 95% CI 2-sided [-0.87 to 1.09]

40. Secondary Outcome: Change From Double-Blind Baseline in Physician Global Evaluation of Disease Activity at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 39
Time Frame: DB label Baseline (last value collected prior to Day 1 of tofacitinib administration in OL phase), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 39
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | 0.16 (0.25) | 0.21 (0.24)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | 0.45 (0.32) | -0.14 (0.32)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | 0.10 (0.40) | -0.02 (0.39)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -0.11 (0.34) | 0.15 (0.34)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -0.51 (0.22) | -0.35 (0.23)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -0.32 (0.22) | -0.37 (0.22)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | 0.09 (0.43) | 0.19 (0.47)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -0.11 (0.29) | -0.42 (0.32)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -0.74 (0.17) | -0.92 (0.18)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -0.17 (0.35) | -0.53 (0.37)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -0.79 (0.21) | -0.70 (0.22)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -1.03 (0.20) | -1.09 (0.29)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -1.00 (0.27) | -0.92 (0.39)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 1]; Test type: Other; Difference in LS Mean = -0.05, 95% CI 2-sided [-0.77 to 0.67]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 2]; Test type: Other; Difference in LS Mean = 0.58, 95% CI 2-sided [-0.37 to 1.53]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 3]; Test type: Other; Difference in LS Mean = 0.12, 95% CI 2-sided [-1.06 to 1.30]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 4]; Test type: Other; Difference in LS Mean = -0.26, 95% CI 2-sided [-1.27 to 0.74]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 5]; Test type: Other; Difference in LS Mean = -0.16, 95% CI 2-sided [-0.83 to 0.52]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 6]; Test type: Other; Difference in LS Mean = 0.05, 95% CI 2-sided [-0.61 to 0.71]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 7]; Test type: Other; Difference in LS Mean = -0.10, 95% CI 2-sided [-1.45 to 1.25]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 8]; Test type: Other; Difference in LS Mean = 0.31, 95% CI 2-sided [-0.61 to 1.23]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 9]; Test type: Other; Difference in LS Mean = 0.18, 95% CI 2-sided [-0.34 to 0.71]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 10]; Test type: Other; Difference in LS Mean = 0.36, 95% CI 2-sided [-0.74 to 1.46]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 11]; Test type: Other; Difference in LS Mean = -0.09, 95% CI 2-sided [-0.75 to 0.56]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 12]; Test type: Other; Difference in LS Mean = 0.06, 95% CI 2-sided [-0.68 to 0.81]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 13]; Test type: Other; Difference in LS Mean = -0.08, 95% CI 2-sided [-1.10 to 0.94]

41. Secondary Outcome: Change From Open-Label Baseline in ESR at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: ESR was determined using an ESR testing kit.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Millimeter per hour (mm/h)
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Millimeter per hour (mm/h)
  DB Week 4: number analyzed (Participants) | 27 | 31
  DB Week 4 | -32.65 (4.72) | -31.19 (4.49)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | -36.55 (4.38) | -29.32 (4.29)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | -38.30 (4.50) | -31.69 (4.35)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -39.52 (4.06) | -31.02 (4.06)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -41.82 (2.22) | -37.86 (2.32)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -42.25 (2.25) | -40.81 (2.33)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -37.83 (4.07) | -33.51 (4.39)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -37.90 (3.67) | -35.04 (3.91)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -39.36 (4.49) | -28.41 (4.79)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -39.98 (4.12) | -35.70 (4.31)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -47.16 (2.28) | -38.84 (2.34)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -47.16 (2.29) | -42.32 (2.72)
  DB Week 52: number analyzed (Participants) | 6 | 4
  DB Week 52 | -51.46 (1.08) | -50.12 (1.24)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 1]; Test type: Other; Difference in LS Mean = -1.46, 95% CI 2-sided [-14.59 to 11.66]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 2]; Test type: Other; Difference in LS Mean = -7.22, 95% CI 2-sided [-19.62 to 5.17]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 3]; Test type: Other; Difference in LS Mean = -6.61, 95% CI 2-sided [-19.36 to 6.14]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 4]; Test type: Other; Difference in LS Mean = -8.50, 95% CI 2-sided [-20.28 to 3.27]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 5]; Test type: Other; Difference in LS Mean = -3.95, 95% CI 2-sided [-10.53 to 2.62]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 6]; Test type: Other; Difference in LS Mean = -1.44, 95% CI 2-sided [-8.09 to 5.21]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 7]; Test type: Other; Difference in LS Mean = -4.32, 95% CI 2-sided [-16.67 to 8.03]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 8]; Test type: Other; Difference in LS Mean = -2.86, 95% CI 2-sided [-13.97 to 8.25]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 9]; Test type: Other; Difference in LS Mean = -10.95, 95% CI 2-sided [-24.63 to 2.73]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 10]; Test type: Other; Difference in LS Mean = -4.28, 95% CI 2-sided [-16.74 to 8.18]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 11]; Test type: Other; Difference in LS Mean = -8.32, 95% CI 2-sided [-15.20 to -1.43]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 12]; Test type: Other; Difference in LS Mean = -4.84, 95% CI 2-sided [-12.60 to 2.92]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 37, analysis 13]; Test type: Other; Difference in LS Mean = -1.34, 95% CI 2-sided [-5.16 to 2.48]

42. Secondary Outcome: Change From Double-Blind Baseline in ESR at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: ESR was determined using an ESR testing kit.
Time Frame: DB Baseline (values at randomization), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Millimeter/ hour (mm/h)
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Millimeter/ hour (mm/h)
  DB Week 4: number analyzed (Participants) | 27 | 30
  DB Week 4 | 3.35 (3.71) | 9.41 (3.50)
  DB Week 8: number analyzed (Participants) | 25 | 24
  DB Week 8 | 1.94 (3.97) | 12.39 (3.93)
  DB Week 12: number analyzed (Participants) | 21 | 22
  DB Week 12 | 1.42 (4.53) | 12.28 (4.40)
  DB Week 16: number analyzed (Participants) | 21 | 19
  DB Week 16 | 0.45 (4.32) | 13.59 (4.35)
  DB Week 20: number analyzed (Participants) | 19 | 14
  DB Week 20 | -2.04 (2.17) | 4.98 (2.31)
  DB Week 24: number analyzed (Participants) | 18 | 14
  DB Week 24 | -2.51 (2.14) | 2.01 (2.28)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | 1.73 (4.19) | 11.08 (4.55)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | 2.01 (3.78) | 8.77 (4.05)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | 0.88 (4.83) | 16.37 (5.17)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | 0.34 (4.25) | 8.33 (4.47)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -7.05 (2.34) | 3.44 (2.41)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -8.07 (2.38) | -2.14 (2.96)
  DB Week 52: number analyzed (Participants) | 6 | 4
  DB Week 52 | -11.70 (1.39) | -9.14 (1.73)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 1]; Test type: Other; Difference in LS Mean = -6.05, 95% CI 2-sided [-16.30 to 4.19]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 2]; Test type: Other; Difference in LS Mean = -10.46, 95% CI 2-sided [-21.68 to 0.77]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 3]; Test type: Other; Difference in LS Mean = -10.86, 95% CI 2-sided [-23.75 to 2.03]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 4]; Test type: Other; Difference in LS Mean = -13.15, 95% CI 2-sided [-25.83 to -0.46]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 5]; Test type: Other; Difference in LS Mean = -7.02, 95% CI 2-sided [-13.56 to -0.47]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 6]; Test type: Other; Difference in LS Mean = -4.53, 95% CI 2-sided [-11.00 to 1.95]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 7]; Test type: Other; Difference in LS Mean = -9.35, 95% CI 2-sided [-22.24 to 3.54]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 8]; Test type: Other; Difference in LS Mean = -6.75, 95% CI 2-sided [-18.34 to 4.83]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 9]; Test type: Other; Difference in LS Mean = -15.49, 95% CI 2-sided [-30.36 to -0.63]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 10]; Test type: Other; Difference in LS Mean = -7.99, 95% CI 2-sided [-21.00 to 5.03]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 11]; Test type: Other; Difference in LS Mean = -10.49, 95% CI 2-sided [-17.67 to -3.31]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 12]; Test type: Other; Difference in LS Mean = -5.93, 95% CI 2-sided [-13.53 to 1.67]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 19, analysis 13]; Test type: Other; Difference in LS Mean = -2.57, 95% CI 2-sided [-6.37 to 1.24]

43. Secondary Outcome: Change From Open-Label Baseline in CHAQ -Parental Evaluation of Overall Well-being at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: The CHAQ, derived from the adult health assessment questionnaire, comprised of two indices disability and discomfort, and parent global assessment of overall well-being. For assessment of overall well-being, the parent/legal guardian/participant were required to rate the overall well-being by entering a number from 0 to 10 (in 0.5 increments), on a 21-circle VAS where '0'= very well' and '10= very poorly, where higher scores indicated worse condition.
Time Frame: as for outcome 39
Population: as for outcome 39
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 30
  DB Week 4 | -4.31 (0.37) | -5.52 (0.34)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | -4.56 (0.36) | -5.38 (0.35)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | -4.97 (0.34) | -5.28 (0.33)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | -4.88 (0.29) | -5.46 (0.29)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | -5.19 (0.32) | -5.36 (0.34)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | -4.97 (0.29) | -5.62 (0.30)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -5.08 (0.44) | -5.00 (0.48)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -5.63 (0.18) | -5.55 (0.20)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -5.81 (0.18) | -5.87 (0.21)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -5.98 (0.16) | -5.94 (0.18)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -5.95 (0.21) | -5.79 (0.23)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -5.45 (0.31) | -5.30 (0.57)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -6.06 (0.25) | -5.98 (0.43)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 1]; Test type: Other; Difference in LS Mean = 0.51, 95% CI 2-sided [0.20 to 2.22]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 2]; Test type: Other; Difference in LS Mean = 0.82, 95% CI 2-sided [-0.20 to 1.85]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 3]; Test type: Other; Difference in LS Mean = 0.31, 95% CI 2-sided [-0.65 to 1.27]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 4]; Test type: Other; Difference in LS Mean = 0.57, 95% CI 2-sided [-0.26 to 1.41]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 5]; Test type: Other; Difference in LS Mean = 0.16, 95% CI 2-sided [-0.78 to 1.10]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 6]; Test type: Other; Difference in LS Mean = 0.66, 95% CI 2-sided [-0.18 to 1.49]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 7]; Test type: Other; Difference in LS Mean = -0.08, 95% CI 2-sided [-1.43 to 1.27]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 8]; Test type: Other; Difference in LS Mean = -0.07, 95% CI 2-sided [-0.65 to 0.50]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 9]; Test type: Other; Difference in LS Mean = 0.06, 95% CI 2-sided [-0.51 to 0.63]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 10]; Test type: Other; Difference in LS Mean = -0.04, 95% CI 2-sided [-0.55 to 0.47]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 11]; Test type: Other; Difference in LS Mean = -0.16, 95% CI 2-sided [-0.82 to 0.50]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 12]; Test type: Other; Difference in LS Mean = -0.14, 95% CI 2-sided [-1.51 to 1.22]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; [analysis description as in outcome 33, analysis 13]; Test type: Other; Difference in LS Mean = -0.08, 95% CI 2-sided [-1.05 to 0.88]

44. Secondary Outcome: Change From Double-Blind Baseline in CHAQ -Parental Evaluation of Overall Well-being at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: The CHAQ, derived from the adult health assessment questionnaire, comprised of two indices disability and discomfort, and parent global assessment of overall well-being. For assessment of overall well-being, the parent/legal guardian/participant were required to rate the overall well-being by entering a number from 0 to 10 (in 0.5 increments), on a 21-circle VAS where '0'= very well' and '10=very poorly.
Time Frame: DB Baseline (value at randomization), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 39
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 30
  DB Week 4 | 0.46 (0.28) | -0.03 (0.27)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | 0.60 (0.38) | 0.12 (0.38)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | 0.25 (0.36) | 0.22 (0.35)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | 0.27 (0.31) | 0.04 (0.31)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | 0.14 (0.37) | 0.05 (0.38)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | 0.14 (0.29) | -0.14 (0.30)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | 0.54 (0.52) | 0.52 (0.56)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -0.32 (0.24) | -0.34 (0.25)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -0.56 (0.21) | -0.63 (0.22)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -0.72 (0.19) | -0.78 (0.20)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -0.65 (0.24) | -0.54 (0.25)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -0.16 (0.36) | -0.37 (0.53)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -0.82 (0.26) | -0.87 (0.38)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 4: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.49, 95% CI 2-sided [-0.32 to 1.30]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 8: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.48, 95% CI 2-sided [-0.64 to 1.61]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 12: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.03, 95% CI 2-sided [-1.02 to 1.07]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 16: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.23, 95% CI 2-sided [-0.69 to 1.14]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 20: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.09, 95% CI 2-sided [-1.05 to 1.22]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.28, 95% CI 2-sided [-0.60 to 1.16]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 28: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.02, 95% CI 2-sided [-1.60 to 1.64]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 32: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.02, 95% CI 2-sided [-1.60 to 1.64]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 36: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.07, 95% CI 2-sided [-0.58 to 0.73]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 40: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.06, 95% CI 2-sided [-0.53 to 0.65]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 44: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.12, 95% CI 2-sided [-0.87 to 0.64]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.21, 95% CI 2-sided [-1.13 to 1.54]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB at Week 52: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.05, 95% CI 2-sided [-1.00 to 1.11]

45. Secondary Outcome: Change From Open-Label Baseline in Child Health Questionnaire (CHQ) Responses at End of Open-Label Phase Part 1
Description: The CHQ is a validated general pediatric quality of life instrument. The CHQ assessed for 14 physical and psychosocial domains: general health perceptions (global health perception), physical functioning, role/social physical functioning, bodily pain, role/social emotional functioning, role/social behavioral functioning, parent/legal guardian/adult caregiver impact-time, parent/legal guardian/adult caregiver impact-emotional, self-esteem, mental health, behavior, family activities, family cohesion, and change in health. The response options for the CHQ are ordinal scales that vary by the item. Each item consisted of 4-6 response options. The CHQ score was determined based on the parent/legal guardian/adult caregiver's questionnaire responses. Range on subscales and the overall scale is 0 to 100, where 0 is the worst possible health state and 100 the best possible health state.
Time Frame: OL Baseline up to 16 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Units on a scale
  Global Health Subscale Standardized Score: number analyzed (Participants) | 85
  Global Health Subscale Standardized Score | 26.12 (29.10)
  Physical Functioning Subscale Standardized Score: number analyzed (Participants) | 85
  Physical Functioning Subscale Standardized Score | 28.95 (33.79)
  Social Limitations: Emotional Subscale Standardized Score: number analyzed (Participants) | 84
  Social Limitations: Emotional Subscale Standardized Score | 27.51 (38.39)
  Social Limitations: Physical Subscale Standardized Score: number analyzed (Participants) | 84
  Social Limitations: Physical Subscale Standardized Score | 31.15 (42.96)
  Bodily Pain Subscale Standardized Score: number analyzed (Participants) | 85
  Bodily Pain Subscale Standardized Score | 32.00 (26.67)
  Behavior Subscale Standardized Score: number analyzed (Participants) | 85
  Behavior Subscale Standardized Score | 10.98 (17.14)
  Global Behavior Subscale Standardized Score: number analyzed (Participants) | 85
  Global Behavior Subscale Standardized Score | 11.18 (27.75)
  Mental Health Subscale Standardized Score: number analyzed (Participants) | 84
  Mental Health Subscale Standardized Score | 13.33 (20.20)
  Self Esteem Subscale Standardized Score: number analyzed (Participants) | 83
  Self Esteem Subscale Standardized Score | 7.68 (21.29)
  General Health Subscale Standardized Score: number analyzed (Participants) | 85
  General Health Subscale Standardized Score | 8.37 (13.93)
  Change in Health Subscale Score: number analyzed (Participants) | 85
  Change in Health Subscale Score | 1.28 (1.10)
  Emotional Impact on Parent Subscale Standardized Score: number analyzed (Participants) | 85
  Emotional Impact on Parent Subscale Standardized Score | 12.75 (26.43)
  Time Impact on Parent Subscale Standardized Score: number analyzed (Participants) | 84
  Time Impact on Parent Subscale Standardized Score | 14.81 (28.62)
  Family Activities Subscale Standardized Score: number analyzed (Participants) | 84
  Family Activities Subscale Standardized Score | 74.03 (22.41)
  Family Cohesion Subscale Standardized Score: number analyzed (Participants) | 84
  Family Cohesion Subscale Standardized Score | 8.10 (22.67)

46. Secondary Outcome: Change From Open-Label Baseline in CHQ Responses at End of Open-Label Phase Part 2
Description: as for outcome 45
Time Frame: Baseline (last value collected prior to Day 1 of tofacitinib administration in OL phase) up to 24 weeks
Population: OLPT2 analysis set included all participants who were enrolled into the OL part 2 phase of the study and received at least one dose of investigational product in part 2. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 29
Units on a scale
  Global Health Standardized Score | 25.52 (35.46)
  Physical Functioning Standardized Score | 33.33 (31.29)
  Social Limitations: Emotional Score: number analyzed (Participants) | 28
  Social Limitations: Emotional Score | 28.17 (43.98)
  Social Limitations: Physical Score: number analyzed (Participants) | 28
  Social Limitations: Physical Score | 38.10 (42.28)
  Bodily Pain Standardized Score | 34.48 (26.80)
  Behavior Standardized Score | 13.02 (21.14)
  Global Behavior Standardized Score | 10.00 (34.10)
  Mental Health Standardized Score: number analyzed (Participants) | 28
  Mental Health Standardized Score | 18.04 (21.01)
  Self Esteem Standardized Score: number analyzed (Participants) | 27
  Self Esteem Standardized Score | 8.30 (34.18)
  General Health Standardized Score: number analyzed (Participants) | 28
  General Health Standardized Score | 8.18 (15.94)
  Change in Health Subscale Score: number analyzed (Participants) | 28
  Change in Health Subscale Score | 1.54 (1.23)
  Emotional Impact on Parent Standardized Score: number analyzed (Participants) | 28
  Emotional Impact on Parent Standardized Score | 22.92 (36.33)
  Time Impact on Parent Standardized Score: number analyzed (Participants) | 27
  Time Impact on Parent Standardized Score | 34.57 (25.66)
  Family Activities Standardized Score: number analyzed (Participants) | 27
  Family Activities Standardized Score | 27.62 (25.87)
  Family Cohesion Standardized Score: number analyzed (Participants) | 27
  Family Cohesion Standardized Score | 10.00 (23.25)

47. Secondary Outcome: Change From Double-Blind Baseline in CHQ Responses at DB Weeks 24, 48: Double-Blind Phase
Description: as for outcome 45
Time Frame: DB Baseline (values at randomization), DB Weeks 24, 48
Population: as for outcome 36
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 17 | 15
Units on a scale
  CHQ01-Global Health Subscale Standardized Score: DB Week 24 | 4.02 (4.71) | -1.98 (5.02)
  CHQ01-Global Health Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Global Health Subscale Standardized Score: DB Week 48 | 4.09 (3.93) | 1.24 (4.49)
  CHQ01-Physical Functioning Subscale Standardized Score: DB Week 24 | 2.51 (3.86) | 6.70 (3.99)
  CHQ01-Physical Functioning Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Physical Functioning Subscale Standardized Score: DB Week 48 | 5.24 (9.13) | 2.93 (14.02)
  CHQ01-Social Limitations: Emotional Subscale Standardized Score: DB Week 24 | 2.62 (4.00) | 8.09 (4.18)
  CHQ01-Social Limitations: Emotional Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Social Limitations: Emotional Subscale Standardized Score: DB Week 48 | 6.09 (7.69) | -0.73 (10.33)
  CHQ01-Social Limitations: Physical Subscale Standardized Score: DB Week 24 | 2.75 (4.27) | 8.98 (4.54)
  CHQ01-Social Limitations: Physical Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Social Limitations: Physical Subscale Standardized Score: DB Week 48 | 3.45 (13.33) | -7.64 (20.06)
  CHQ01-Bodily Pain Subscale Standardized Score: DB Week 24 | -1.61 (4.19) | -0.16 (4.41)
  CHQ01-Bodily Pain Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Bodily Pain Subscale Standardized Score: DB Week 48 | -2.72 (10.19) | -19.92 (13.98)
  CHQ01-Behavior Subscale Standardized Score: DB Week 24 | 2.33 (2.68) | 7.48 (2.87)
  CHQ01-Behavior Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Behavior Subscale Standardized Score: DB Week 48 | -4.50 (4.97) | 10.53 (5.35)
  CHQ01-Global Behavior Subscale Standardized Score: DB Week 24 | 4.17 (3.89) | 9.48 (4.13)
  CHQ01-Global Behavior Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Global Behavior Subscale Standardized Score: DB Week 48 | 5.90 (4.00) | 13.14 (4.54)
  CHQ01-Mental Health Subscale Standardized Score: DB Week 24 | 6.59 (3.56) | 2.14 (3.78)
  CHQ01-Mental Health Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Mental Health Subscale Standardized Score: DB Week 48 | 0.79 (4.98) | 8.26 (5.71)
  CHQ01-Self Esteem Subscale Standardized Score: DB Week 24 | 6.68 (3.05) | 6.69 (3.24)
  CHQ01-Self Esteem Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Self Esteem Subscale Standardized Score: DB Week 48 | 3.05 (7.24) | 10.64 (8.04)
  CHQ01-General Health Subscale Standardized Score: DB Week 24 | 5.02 (3.21) | 0.03 (3.42)
  CHQ01-General Health Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-General Health Subscale Standardized Score: DB Week 48 | 9.59 (5.20) | 10.60 (5.92)
  CHQ01-Change in Health Subscale Score: DB Week 24 | 0.45 (0.12) | 0.48 (0.13)
  CHQ01-Change in Health Subscale Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Change in Health Subscale Score: DB Week 48 | 0.64 (0.32) | 0.16 (0.35)
  CHQ01-Emotion al Impact on Parent Subscale Standardized Score: DB Week 24 | 15.00 (4.28) | 12.75 (4.53)
  CHQ01-Emotion al Impact on Parent Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Emotion al Impact on Parent Subscale Standardized Score: DB Week 48 | 7.15 (10.25) | 32.22 (11.79)
  CHQ01-Time Impact on Parent Subscale Standardized Score: DB Week 24 | 7.53 (5.10) | 5.66 (5.25)
  CHQ01-Time Impact on Parent Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Time Impact on Parent Subscale Standardized Score: DB Week 48 | 11.60 (8.94) | 20.79 (14.05)
  CHQ01-Family Activities Subscale Standardized Score: DB Week 24 | 5.71 (2.96) | 9.68 (3.13)
  CHQ01-Family Activities Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Family Activities Subscale Standardized Score: DB Week 48 | 6.65 (5.73) | 15.95 (7.16)
  CHQ01-Family Cohesion Subscale Standardized Score: DB Week 24 | 2.84 (3.71) | 6.36 (3.96)
  CHQ01-Family Cohesion Subscale Standardized Score: DB Week 48: number analyzed (Participants) | 5 | 4
  CHQ01-Family Cohesion Subscale Standardized Score: DB Week 48 | -12.24 (13.08) | 8.18 (15.58)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Global Health Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 6.00, 95% CI 2-sided [-8.35 to 20.36]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Global Health Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 2.85, 95% CI 2-sided [-12.43 to 18.14]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Physical Functioning Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -4.19, 95% CI 2-sided [-15.78 to 7.40]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Physical Functioning Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 2.31, 95% CI 2-sided [-37.06 to 41.68]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Social Limitations: Emotional Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -5.47, 95% CI 2-sided [-17.37 to 6.43]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Social Limitations: Emotional Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 6.82, 95% CI 2-sided [-20.92 to 34.57]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Social Limitations: Physical Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -6.22, 95% CI 2-sided [-18.95 to 6.50]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Social Limitations: Physical Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 11.09, 95% CI 2-sided [-46.24 to 68.42]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Bodily Pain Subscale Standardized Score: DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -1.45, 95% CI 2-sided [-13.97 to 11.06]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Bodily Pain Subscale Standardized Score: DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 17.20, 95% CI 2-sided [-28.01 to 62.41]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Behavior Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -5.15, 95% CI 2-sided [-13.24 to 2.93]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Behavior Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -15.03, 95% CI 2-sided [-33.12 to 3.06]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Global Behavior Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -5.32, 95% CI 2-sided [-16.92 to 6.29]
Statistical Analysis 14: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Global Behavior Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -7.24, 95% CI 2-sided [-20.35 to 5.87]
Statistical Analysis 15: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Mental Health Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 4.44, 95% CI 2-sided [-6.18 to 15.07]
Statistical Analysis 16: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Mental Health Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -7.46, 95% CI 2-sided [-24.37 to 9.45]
Statistical Analysis 17: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Self Esteem Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.01, 95% CI 2-sided [-9.14 to 9.13]
Statistical Analysis 18: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Self Esteem Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -7.59, 95% CI 2-sided [-33.87 to 18.70]
Statistical Analysis 19: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-General Health Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 4.98, 95% CI 2-sided [-4.81 to 14.77]
Statistical Analysis 20: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-General Health Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -1.02, 95% CI 2-sided [-20.31 to 18.28]
Statistical Analysis 21: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Change in Health Subscale Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.03, 95% CI 2-sided [-0.40 to 0.33]
Statistical Analysis 22: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Change in Health Subscale Score; DB Week48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.48, 95% CI 2-sided [-0.68 to 1.65]
Statistical Analysis 23: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Emotional Impact on Parent Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 2.25, 95% CI 2-sided [-10.59 to 15.10]
Statistical Analysis 24: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Emotional Impact on Parent Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -25.07, 95% CI 2-sided [-60.96 to 10.82]
Statistical Analysis 25: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Time Impact on Parent Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 1.87, 95% CI 2-sided [-13.55 to 17.29]
Statistical Analysis 26: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Time Impact on Parent Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -9.19, 95% CI 2-sided [-48.91 to 30.53]
Statistical Analysis 27: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Family Activities Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -3.97, 95% CI 2-sided [-12.84 to 4.90]
Statistical Analysis 28: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Family Activities Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -9.30, 95% CI 2-sided [-32.35 to 13.75]
Statistical Analysis 29: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Family Cohesion Subscale Standardized Score; DB Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -3.52, 95% CI 2-sided [-14.84 to 7.81]
Statistical Analysis 30: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHQ01-Family Cohesion Subscale Standardized Score; DB Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -20.42, 95% CI 2-sided [-79.03 to 38.18]

48. Secondary Outcome: Change From Open-Label Baseline in CHAQ-Discomfort Index at Part 1 Day 7, Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: For the assessment of discomfort, the parent/legal guardian or adult caregiver who interacted daily with the participant were required to rate the overall pain the participant had due to illness by entering a number from 0 to 10 (in 0.5 increments), with '0' as 'no pain' and '10' as 'very severe pain' on a 21-circle VAS, where higher scores indicated more severe pain.
Time Frame: Baseline (last value collected prior to Day 1 of tofacitinib administration in OL phase) Part 1 Day 7, Weeks 2, 4, 8, 12, 16
Population: OLPT1 consisted of all participants who were enrolled into the OL part 1 and received at least one dose of investigational product in part 1. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Units on a scale
  Part 1 Day 7: number analyzed (Participants) | 99
  Part 1 Day 7 | -1.20 (1.77)
  Part 1 Week 2: number analyzed (Participants) | 98
  Part 1 Week 2 | -1.87 (2.07)
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | -2.57 (2.14)
  Part 1 Week 8: number analyzed (Participants) | 82
  Part 1 Week 8 | -3.30 (2.45)
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | -3.57 (2.50)
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | -3.69 (2.28)

49. Secondary Outcome: Change From Open-label Baseline in CHAQ-Discomfort Index at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: For the assessment of discomfort, the parent/legal guardian or adult caregiver who interacted daily with the participant were required to rate the overall pain the participant had due to illness by entering a number from 0 to 10 (in 0.5 increments), with '0' as 'no pain' and '10' as 'very severe pain' on a 21-circle VAS, where higher scores indicated more pain.
Time Frame: Baseline (last value collected prior to Day 1 of tofacitinib administration in OL phase) Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: OLPT2 consisted of all participants who were enrolled into the OL part 2 and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Units on a scale
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | -4.23 (3.14)
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | -4.38 (2.95)
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | -4.42 (3.26)
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | -4.48 (2.88)
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | -5.15 (3.52)
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | -6.00 (1.73)

50. Secondary Outcome: Change From Double-Blind Baseline in CHAQ-Discomfort Index at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 48
Time Frame: DB Baseline (value at randomization), DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Units on a scale
  DB Week 4: number analyzed (Participants) | 27 | 30
  DB Week 4 | 0.13 (0.28) | 0.37 (0.26)
  DB Week 8: number analyzed (Participants) | 25 | 25
  DB Week 8 | 0.56 (0.36) | 0.02 (0.35)
  DB Week 12: number analyzed (Participants) | 21 | 23
  DB Week 12 | 0.04 (0.34) | 0.09 (0.32)
  DB Week 16: number analyzed (Participants) | 21 | 20
  DB Week 16 | 0.44 (0.36) | -0.11 (0.35)
  DB Week 20: number analyzed (Participants) | 19 | 15
  DB Week 20 | 0.09 (0.40) | -0.14 (0.42)
  DB Week 24: number analyzed (Participants) | 18 | 15
  DB Week 24 | 0.07 (0.27) | -0.25 (0.28)
  DB Week 28: number analyzed (Participants) | 17 | 12
  DB Week 28 | -0.03 (0.47) | 0.39 (0.51)
  DB Week 32: number analyzed (Participants) | 13 | 10
  DB Week 32 | -0.31 (0.39) | 0.01 (0.42)
  DB Week 36: number analyzed (Participants) | 13 | 10
  DB Week 36 | -0.55 (0.34) | -0.24 (0.37)
  DB Week 40: number analyzed (Participants) | 11 | 9
  DB Week 40 | -0.76 (0.20) | -0.83 (0.21)
  DB Week 44: number analyzed (Participants) | 10 | 9
  DB Week 44 | -1.09 (0.23) | -0.79 (0.24)
  DB Week 48: number analyzed (Participants) | 8 | 5
  DB Week 48 | -0.19 (0.49) | -0.43 (0.79)
  DB Week 52: number analyzed (Participants) | 6 | 5
  DB Week 52 | -0.85 (0.21) | -0.76 (0.34)
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 4: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.24, 95% CI 2-sided [-1.02 to 0.54]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 8: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.54, 95% CI 2-sided [-0.49 to 1.57]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 12: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.47, 95% CI 2-sided [-1.01 to 0.90]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 16: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.55, 95% CI 2-sided [-0.49 to 1.58]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 20: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.23, 95% CI 2-sided [-0.98 to 1.45]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 24: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.32, 95% CI 2-sided [-0.51 to 1.14]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 28: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.42, 95% CI 2-sided [-1.87 to 1.03]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 32: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.33, 95% CI 2-sided [-1.53 to 0.88]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 36: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.31, 95% CI 2-sided [-1.36 to 0.74]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 40: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.07, 95% CI 2-sided [-0.55 to 0.69]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 44: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.31, 95% CI 2-sided [-1.01 to 0.39]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 48: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = 0.23, 95% CI 2-sided [-1.45 to 1.92]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; CHAQ-Discomfort Index at Week 52: Analysis performed using MMRM which included the fixed effect of treatment, visit, treatment by visit interaction, Double-Blind baseline value, and Double-Blind baseline value by visit interaction; Test type: Other; Difference in LS Mean = -0.09, 95% CI 2-sided [-0.87 to 0.69]

51. Secondary Outcome: Percentage of Participants With Minimum Disease Activity Calculated From JADAS-27 CRP Score at Part 1 Day 7, Weeks 2, 4, 8, 12 and 16: Open-Label Phase Part 1
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 CRP score were determined based on four components: Physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 (very well) to 10 (very poor), CRP (value normalized to 0 to 10 scale, where higher scores indicated more inflammation) and number of joints with active disease (27 joint assessment ranging from 0 to 27, where higher scores indicated more disease activity). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57, where higher scores indicated more disease activity. For participants with polyarthritis (>4 active joints) minimal disease activity was defined as a JADAS-27 CRP score of: <= 3.8. For participants with oligoarthritis (<= 4 active joints) minimal disease activity was defined as a JADAS-27 CRP score of <=2.
Time Frame: Part 1 Day 7, Part 1 Weeks 2, 4, 8, 12 and 16
Population: OLPT1 consisted of all participants who were enrolled into the OL part 1 and received at least one dose of investigational product in part 1. All participants reported under "Number of participants analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed": participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of participants
  Part 1 Day 7: number analyzed (Participants) | 97
  Part 1 Day 7 | 3.09 [0 to 6.54]
  Part 1 Week 2: number analyzed (Participants) | 96
  Part 1 Week 2 | 5.21 [0.76 to 9.65]
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | 6.19 [1.39 to 10.98]
  Part 1 Week 8: number analyzed (Participants) | 80
  Part 1 Week 8 | 13.75 [6.20 to 21.30]
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | 13.64 [3.50 to 23.78]
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | 25.00 [7.68 to 42.32]

52. Secondary Outcome: Percentage of Participants With Minimum Disease Activity Calculated From JADAS-27 ESR Score at Part 1 Day 7, Weeks 2, 4, 8, 12 and 16: Open-label Phase Part 1
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 ESR score were determined based on four components: Physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 (very well) to 10 (very poor), ESR (value normalized to 0 to 10 scale, where higher scores indicated more inflammation) and number of joints with active disease (27 joint assessment ranging from 0 to 27, where higher scores indicated more disease activity). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57, where higher scores indicated more disease activity. For participants with polyarthritis (>4 active joints) minimal disease activity was defined as a JADAS-27 ESR score of: <= 3.8. For participants with oligoarthritis (<= 4 active joints) minimal disease activity was defined as a JADAS-27 ESR score of <=2.
Time Frame: Part 1 Day 7, Weeks 2, 4, 8, 12 and 16
Population: OLPT1 consisted of all participants who were enrolled into the OL part 1 and received at least one dose of investigational product in part 1. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed": participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of participants
  Part 1 Day 7: number analyzed (Participants) | 98
  Part 1 Day 7 | 1.02 [0 to 3.01]
  Part 1 Week 2: number analyzed (Participants) | 98
  Part 1 Week 2 | 4.08 [0.16 to 8.00]
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | 7.22 [2.07 to 12.37]
  Part 1 Week 8: number analyzed (Participants) | 81
  Part 1 Week 8 | 14.81 [7.08 to 22.55]
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | 15.91 [5.10 to 26.72]
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | 20.83 [4.59 to 37.08]

53. Secondary Outcome: Percentage of Participants With Minimum Disease Activity Calculated From JADAS-27 CRP Score at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 51
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: OLPT2 consisted of all participants who were enrolled into the OL part 2 and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number analyzed": participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | 36.00 [22.70 to 49.30]
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | 30.00 [15.80 to 44.20]
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | 32.26 [15.80 to 48.71]
  Part 2 Week 16: number analyzed (Participants) | 22
  Part 2 Week 16 | 36.36 [16.26 to 56.47]
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | 53.85 [26.75 to 80.95]
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | 33.33 [0 to 86.68]

54. Secondary Outcome: Percentage of Participants With Minimum Disease Activity Calculated From JADAS-27 ESR Score at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 52
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 53
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | 32.00 [19.07 to 44.93]
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | 27.50 [13.66 to 41.34]
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | 29.03 [13.05 to 45.01]
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | 34.78 [15.32 to 54.25]
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | 53.85 [26.75 to 80.95]
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | 33.33 [0 to 86.68]

55. Secondary Outcome: Percentage of Participants With Inactive Disease Status Calculated From JADAS-27 CRP Score at Part 1 Day 7, Weeks 2, 4, 8, 12 and 16: Open-label Phase Part 1
Description: JADAS-27 is a validated composite disease activity measure for JIA. Score were determined based on four components:Physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 (very well) to 10 (very poor), CRP (value normalized to 0 to 10 scale, where higher scores:more inflammation) and number of joints with active disease (27 joint assessment ranging from 0 to 27,where higher scores:more disease activity). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57,where higher scores:more disease activity.Inactive disease activity based on JADAS-27 CRP score was defined as: For participants with polyarthritis (>4 active joints) inactive disease activity was defined as a JADAS-27 CRP score of:<=1.For participants with oligoarthritis (<=4 active joints) inactive disease activity was defined as a JADAS-27 CRP score of <=1.
Time Frame: Part 1 Day 7, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 52
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of Participants
  Part 1 Day 7: number analyzed (Participants) | 97
  Part 1 Day 7 | 0 [0 to 0]
  Part 1 Week 2: number analyzed (Participants) | 96
  Part 1 Week 2 | 3.13 [0 to 6.61]
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | 3.09 [0 to 6.54]
  Part 1 Week 8: number analyzed (Participants) | 80
  Part 1 Week 8 | 5.00 [0.22 to 9.78]
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | 4.55 [0 to 10.70]
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | 4.17 [0 to 12.16]

56. Secondary Outcome: Percentage of Participants With Inactive Disease Status Calculated From JADAS-27 ESR Score at Part 1 Day 7, Weeks 2, 4, 8, 12 and 16: Open-Label Phase Part 1
Description: JADAS-27 is a validated composite disease activity measure for JIA. Score were determined based on four components:physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity);parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 (very well) to 10 (very poor), ESR (value normalized to 0 to 10 scale, where higher scores:more inflammation and number of joints with active disease (27 joint assessment ranging from 0 to 27, where higher scores:more disease activity). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57, where higher scores:more disease activity. Inactive Disease activity based on JADAS-27 ESR score was defined as for participants with polyarthritis(>4 active joints) inactive disease activity was defined as a JADAS-27 ESR score of:<=1. For participants with oligoarthritis (<=4 active joints) inactive disease activity was defined as a JADAS-27 ESR score of <=1.
Time Frame: Part 1 Day 7, Weeks 2, 4, 8, 12 and 16
Population: OLPT1 consisted of all participants who were enrolled into the OL part 1 and received at least one dose of investigational product in part 1. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed": participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of Participants
  Part 1 Day 7: number analyzed (Participants) | 98
  Part 1 Day 7 | 0 [0 to 0]
  Part 1 Week 2: number analyzed (Participants) | 98
  Part 1 Week 2 | 2.04 [0 to 4.84]
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | 1.03 [0 to 3.04]
  Part 1 Week 8: number analyzed (Participants) | 81
  Part 1 Week 8 | 3.70 [0 to 7.82]
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | 6.82 [0 to 14.27]
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | 4.17 [0 to 12.16]

57. Secondary Outcome: Percentage of Participants With Inactive Disease Status Calculated From JADAS-27 CRP Score at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: JADAS-27 is a validated composite disease activity measure for JIA.Score were determined based on four components:physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity);parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 (very well) to 10 (very poor), CRP (value normalized to 0 to 10 scale, where higher scores: more inflammation) and number of joints with active disease (27 joint assessment ranging from 0 to 27,where higher scores:more disease activity). The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57,where higher scores: more disease activity.Inactive disease activity based on JADAS-27 CRP score was defined as: For participants with polyarthritis (>4 active joints) inactive disease activity was defined as a JADAS-27 CRP score of:<=1.For participants with oligoarthritis (<=4 active joints) inactive disease activity was defined as a JADAS-27 CRP score of <=1.
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: OLPT2 consisted of all participants who were enrolled into the OL part 2 and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed": participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of Participants
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | 16.00 [5.84 to 26.16]
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | 20.00 [7.60 to 32.40]
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | 9.68 [0 to 20.09]
  Part 2 Week 16: number analyzed (Participants) | 22
  Part 2 Week 16 | 18.18 [2.06 to 34.30]
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | 38.46 [12.01 to 64.91]
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | 33.33 [0 to 86.68]

58. Secondary Outcome: Percentage of Participants With Inactive Disease Status Calculated From JADAS-27 ESR Score at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: as for outcome 56
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of Participants
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | 16.00 [5.84 to 26.16]
  Part 2 Week 8: number analyzed (Participants) | 40
  Part 2 Week 8 | 17.50 [5.72 to 29.28]
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | 9.68 [0 to 20.09]
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | 17.39 [1.90 to 32.88]
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | 46.15 [19.05 to 73.25]
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | 33.33 [0 to 86.68]

59. Secondary Outcome: Percentage of Participants With Minimum Disease Activity Calculated From JADAS-27 CRP Score at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 51
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage of Participants
  DB Week 4 | 21.43 | 51.61
  DB Week 8 | 25.00 | 48.39
  DB Week 12 | 32.14 | 32.26
  DB Week 16 | 35.71 | 29.03
  DB Week 20 | 35.71 | 22.58
  DB Week 24 | 35.71 | 35.48
  DB Week 28 | 35.71 | 32.26
  DB Week 32 | 28.57 | 22.58
  DB Week 36 | 39.29 | 35.48
  DB Week 40 | 39.29 | 29.03
  DB Week 44 | 46.43 | 25.81
  DB Week 48 | 46.43 | 25.81
  DB Week 52 | 46.43 | 29.03
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4; Test type: Other; Difference in percentage = -30.18, 95% CI 2-sided [-53.43 to -6.94] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8; Test type: Other; Difference in percentage = -23.39, 95% CI 2-sided [-47.19 to 0.42] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12; Test type: Other; Difference in percentage = -0.12, 95% CI 2-sided [-23.99 to 23.76] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16; Test type: Other; Difference in percentage = 6.68, 95% CI 2-sided [-17.20 to 30.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20; Test type: Other; Difference in percentage = 13.13, 95% CI 2-sided [-9.92 to 36.19] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24; Test type: Other; Difference in percentage = 0.23, 95% CI 2-sided [-24.24 to 24.70] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28; Test type: Other; Difference in percentage = 3.46, 95% CI 2-sided [-20.75 to 27.66] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32; Test type: Other; Difference in percentage = 5.99, 95% CI 2-sided [-16.29 to 28.28] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36; Test type: Other; Difference in percentage = 3.80, 95% CI 2-sided [-20.92 to 28.52] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40; Test type: Other; Difference in percentage = 10.25, 95% CI 2-sided [-13.88 to 34.39] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44; Test type: Other; Difference in percentage = 20.62, 95% CI 2-sided [-3.43 to 44.67] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48; Test type: Other; Difference in percentage = 20.62, 95% CI 2-sided [-3.43 to 44.67] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52; Test type: Other; Difference in percentage = 17.40, 95% CI 2-sided [-7.03 to 41.82] — [estimate comment as in outcome 5, analysis 1]

60. Secondary Outcome: Percentage of Participants With Minimum Disease Activity Calculated From JADAS-27 ESR Score at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 52
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage of Participants
  DB Week 4 | 25.00 | 51.61
  DB Week 8 | 25.00 | 45.16
  DB Week 12 | 32.14 | 41.94
  DB Week 16 | 35.71 | 35.48
  DB Week 20 | 39.29 | 29.03
  DB Week 24 | 35.71 | 38.71
  DB Week 28 | 35.71 | 38.71
  DB Week 32 | 28.57 | 35.48
  DB Week 36 | 39.29 | 35.48
  DB Week 40 | 39.29 | 32.26
  DB Week 44 | 50.00 | 32.26
  DB Week 48 | 50.00 | 35.48
  DB Week 52 | 50.00 | 32.26
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4; Test type: Other; Difference in percentage = -26.61, 95% CI 2-sided [-50.42 to -2.81] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8; Test type: Other; Difference in percentage = -20.16, 95% CI 2-sided [-43.91 to 3.59] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12; Test type: Other; Difference in percentage = -9.79, 95% CI 2-sided [-34.31 to 14.72] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16; Test type: Other; Difference in percentage = 0.23, 95% CI 2-sided [-24.24 to 24.70] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20; Test type: Other; Difference in percentage = 10.25, 95% CI 2-sided [-13.88 to 34.39] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24; Test type: Other; Difference in percentage = -3.00, 95% CI 2-sided [-27.67 to 21.68] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28; Test type: Other; Difference in percentage = -3.00, 95% CI 2-sided [-27.67 to 21.68] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32; Test type: Other; Difference in percentage = -6.91, 95% CI 2-sided [-30.65 to 16.83] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36; Test type: Other; Difference in percentage = 3.80, 95% CI 2-sided [-20.92 to 28.52] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40; Test type: Other; Difference in percentage = 7.03, 95% CI 2-sided [-17.43 to 31.48] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44; Test type: Other; Difference in percentage = 17.74, 95% CI 2-sided [-7.03 to 42.52] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48; Test type: Other; Difference in percentage = 14.52, 95% CI 2-sided [-10.52 to 39.55] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52; Test type: Other; Difference in percentage = 17.74, 95% CI 2-sided [-7.03 to 42.52] — [estimate comment as in outcome 5, analysis 1]

61. Secondary Outcome: Percentage of Participants With Inactive Disease Status Calculated From JADAS-27 CRP Score at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-blind Phase
Description: JADAS-27 is a validated composite disease activity measure for JIA.Score were determined based on four components:physician global assessment of disease activity assessed on a VAS of 0 (no activity) to 10 (maximum activity); parent/legal guardian global assessment of well-being (from the CHAQ assessed on a VAS of 0 (very well) to 10 (very poor),CRP (value normalized to 0 to 10 scale, where higher scores:more inflammation) and number of joints with active disease (27 joint assessment ranging from 0 to 27, where higher scores:more disease activity).The overall JADAS-27 score was sum of the 4 components and it ranged from 0 to 57, where higher scores:more disease activity. Inactive disease activity based on JADAS-27 CRP score was defined as: For participants with polyarthritis (>4 active joints) inactive disease activity was defined as a JADAS-27 CRP score of:<=1.For participants with oligoarthritis (<=4 active joints) inactive disease activity was defined as a JADAS-27 CRP score of <=1.
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage of Participants
  DB Week 4 | 10.71 | 25.81
  DB Week 8 | 7.14 | 19.35
  DB Week 12 | 7.14 | 16.13
  DB Week 16 | 14.29 | 9.68
  DB Week 20 | 14.29 | 9.68
  DB Week 24 | 7.14 | 16.13
  DB Week 28 | 10.71 | 22.58
  DB Week 32 | 14.29 | 19.35
  DB Week 36 | 10.71 | 16.13
  DB Week 40 | 14.29 | 25.81
  DB Week 44 | 14.29 | 16.13
  DB Week 48 | 10.71 | 19.35
  DB Week 52 | 14.29 | 19.35
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4; Test type: Other; Difference in percentage = -15.09, 95% CI 2-sided [-34.29 to 4.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8; Test type: Other; Difference in percentage = -12.21, 95% CI 2-sided [-29.08 to 4.65] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12; Test type: Other; Difference in percentage = -8.99, 95% CI 2-sided [-25.07 to 7.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16; Test type: Other; Difference in percentage = 4.61, 95% CI 2-sided [-12.01 to 21.23] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20; Test type: Other; Difference in percentage = 4.61, 95% CI 2-sided [-12.01 to 21.23] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24; Test type: Other; Difference in percentage = -8.99, 95% CI 2-sided [-25.07 to 7.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28; Test type: Other; Difference in percentage = -11.87, 95% CI 2-sided [-30.52 to 6.79] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32; Test type: Other; Difference in percentage = -5.07, 95% CI 2-sided [-24.08 to 13.94] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36; Test type: Other; Difference in percentage = -5.41, 95% CI 2-sided [-22.70 to 11.87] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40; Test type: Other; Difference in percentage = -11.52, 95% CI 2-sided [-31.65 to 8.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44; Test type: Other; Difference in percentage = -1.84, 95% CI 2-sided [-20.16 to 16.48] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48; Test type: Other; Difference in percentage = -8.64, 95% CI 2-sided [-26.66 to 9.38] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52; Test type: Other; Difference in percentage = -5.07, 95% CI 2-sided [-24.08 to 13.94] — [estimate comment as in outcome 5, analysis 1]

62. Secondary Outcome: Percentage of Participants With Inactive Disease Status Calculated From JADAS-27 ESR Score at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 56
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage of Participants
  DB Week 4 | 7.14 | 19.35
  DB Week 8 | 14.29 | 29.03
  DB Week 12 | 14.29 | 22.58
  DB Week 16 | 17.86 | 16.13
  DB Week 20 | 14.29 | 12.90
  DB Week 24 | 10.71 | 16.13
  DB Week 28 | 10.71 | 22.58
  DB Week 32 | 14.29 | 19.35
  DB Week 36 | 10.71 | 19.35
  DB Week 40 | 14.29 | 25.81
  DB Week 44 | 14.29 | 22.58
  DB Week 48 | 14.29 | 22.58
  DB Week 52 | 14.29 | 19.35
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4; Test type: Other; Difference in percentage = -12.21, 95% CI 2-sided [-29.08 to 4.65] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8; Test type: Other; Difference in percentage = -14.75, 95% CI 2-sided [-35.32 to 5.83] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12; Test type: Other; Difference in percentage = -8.29, 95% CI 2-sided [-27.91 to 11.32] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16; Test type: Other; Difference in percentage = 1.73, 95% CI 2-sided [-17.48 to 20.93] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20; Test type: Other; Difference in percentage = 1.38, 95% CI 2-sided [-16.15 to 18.91] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24; Test type: Other; Difference in percentage = -5.41, 95% CI 2-sided [-22.70 to 11.87] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28; Test type: Other; Difference in percentage = -11.87, 95% CI 2-sided [-30.52 to 6.79] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32; Test type: Other; Difference in percentage = -5.07, 95% CI 2-sided [-24.08 to 13.94] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36; Test type: Other; Difference in percentage = -8.64, 95% CI 2-sided [-26.66 to 9.38] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40; Test type: Other; Difference in percentage = -11.52, 95% CI 2-sided [-31.65 to 8.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44; Test type: Other; Difference in percentage = -8.29, 95% CI 2-sided [-27.91 to 11.32] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48; Test type: Other; Difference in percentage = -8.29, 95% CI 2-sided [-27.91 to 11.32] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52; Test type: Other; Difference in percentage = -5.07, 95% CI 2-sided [-24.08 to 13.94] — [estimate comment as in outcome 5, analysis 1]

63. Secondary Outcome: Percentage of Participants With JIA ACR Inactive Disease Status at Part 1 Days 3, 7, Weeks 2, 4, 8, 12, 16: Open-Label Phase Part 1
Description: The ACR clinical inactive disease was defined as follows: no joints with active arthritis; no fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to sJIA; no active uveitis; normal ESR (within normal limits of the method used where tested) or, if elevated, not attributable to JIA; physician global assessment of disease activity score of 'best possible' on the 21-numbered circle VAS scale used (VAS from 0 to 10), higher scores indicated more disease activity; duration of morning stiffness of <=15 minutes. 95% CI was based on normal approximation.
Time Frame: Baseline (last value collected prior to Day 1 of tofacitinib administration in OL phase) Part 1 Days 3, 7, Weeks 2, 4, 8, 12, 16
Population: OLPT1 consisted of all participants who were enrolled into the OL part 1 and received at least one dose of investigational product in part 1. Here "Number analyzed" signifies participants evaluable for specified time points and used for calculating percentages.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID OL Part 1
Number analyzed (Participants) | 100
Percentage of Participants
  Baseline | 0 [0 to 0]
  Part 1 Day 3: number analyzed (Participants) | 96
  Part 1 Day 3 | 0 [0 to 0]
  Part 1 Day 7: number analyzed (Participants) | 99
  Part 1 Day 7 | 0 [0 to 0]
  Part 1 Week 2: number analyzed (Participants) | 99
  Part 1 Week 2 | 2.02 [0 to 4.79]
  Part 1 Week 4: number analyzed (Participants) | 97
  Part 1 Week 4 | 3.09 [0 to 6.54]
  Part 1 Week 8: number analyzed (Participants) | 83
  Part 1 Week 8 | 4.82 [0.21 to 9.43]
  Part 1 Week 12: number analyzed (Participants) | 44
  Part 1 Week 12 | 4.55 [0 to 10.70]
  Part 1 Week 16: number analyzed (Participants) | 24
  Part 1 Week 16 | 4.17 [0 to 12.16]

64. Secondary Outcome: Percentage of Participants With JIA ACR Inactive Disease Status at Part 2 Weeks 4, 8, 12, 16, 20, 24: Open-Label Phase Part 2
Description: The ACR clinical inactive disease was defined as follows: no joints with active arthritis; no fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to sJIA; no active uveitis; normal ESR (within normal limits of the method used where tested) or, if elevated, not attributable to JIA; physician global assessment of disease activity score of 'best possible' on the 21-numbered circle VAS scale used (VAS from 0 to 10), higher scores indicated more disease activity; duration of morning stiffness of <=15 minutes. 95% CI was based on normal approximation. 95% CI was based on normal approximation.
Time Frame: Part 2 Weeks 4, 8, 12, 16, 20, 24
Population: OLPT2 consisted of all participants who were enrolled into the OL part 2 and received at least one dose of investigational product in part 2. All participants reported under 'Number of participants analyzed' contributed data to the table; however, may not have evaluable data for every row. Here "Number analyzed" signifies participants evaluable for specified time points and used for calculating percentages
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5mg BID OL Part 2
Number analyzed (Participants) | 54
Percentage of participants
  Part 2 Week 4: number analyzed (Participants) | 50
  Part 2 Week 4 | 14.00 [4.38 to 23.62]
  Part 2 Week 8: number analyzed (Participants) | 39
  Part 2 Week 8 | 10.26 [0.73 to 19.78]
  Part 2 Week 12: number analyzed (Participants) | 31
  Part 2 Week 12 | 6.45 [0 to 15.10]
  Part 2 Week 16: number analyzed (Participants) | 23
  Part 2 Week 16 | 13.04 [0 to 26.81]
  Part 2 Week 20: number analyzed (Participants) | 13
  Part 2 Week 20 | 15.38 [0 to 35.00]
  Part 2 Week 24: number analyzed (Participants) | 3
  Part 2 Week 24 | 33.33 [0 to 86.68]

65. Secondary Outcome: Percentage of Participants With JIA ACR Inactive Disease Status at DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52: Double-Blind Phase
Description: as for outcome 64
Time Frame: DB Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib 5mg BID DB | Placebo DB
Number analyzed (Participants) | 28 | 31
Percentage of Participants
  DB Week 4 | 7.14 | 16.13
  DB Week 8 | 3.57 | 22.58
  DB Week 12 | 7.14 | 22.58
  DB Week 16 | 3.57 | 16.13
  DB Week 20 | 7.14 | 16.13
  DB Week 24 | 7.14 | 19.35
  DB Week 28 | 10.71 | 19.35
  DB Week 32 | 10.71 | 19.35
  DB Week 36 | 14.29 | 16.13
  DB Week 40 | 17.86 | 22.58
  DB Week 44 | 14.29 | 22.58
  DB Week 48 | 17.86 | 22.58
  DB Week 52 | 21.43 | 19.35
Statistical Analysis 1: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 4; Test type: Other; Difference in percentage = -8.99, 95% CI 2-sided [-25.07 to 7.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 8; Test type: Other; Difference in percentage = -19.01, 95% CI 2-sided [-35.25 to -2.76] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 12; Test type: Other; Difference in percentage = -15.44, 95% CI 2-sided [-32.98 to 2.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 16; Test type: Other; Difference in percentage = -12.56, 95% CI 2-sided [-27.22 to 2.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 20; Test type: Other; Difference in percentage = -8.99, 95% CI 2-sided [-25.07 to 7.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 24; Test type: Other; Difference in percentage = -12.21, 95% CI 2-sided [-29.08 to 4.65] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 28; Test type: Other; Difference in percentage = -8.64, 95% CI 2-sided [-26.66 to 9.38] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 32; Test type: Other; Difference in percentage = -8.64, 95% CI 2-sided [-26.66 to 9.38] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 36; Test type: Other; Difference in percentage = -1.84, 95% CI 2-sided [-20.16 to 16.48] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 40; Test type: Other; Difference in percentage = -4.72, 95% CI 2-sided [-25.17 to 15.72] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 44; Test type: Other; Difference in percentage = -8.29, 95% CI 2-sided [-27.91 to 11.32] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 48; Test type: Other; Difference in percentage = -4.72, 95% CI 2-sided [-25.17 to 15.72] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: Tofacitinib 5mg BID DB vs Placebo DB; DB Week 52; Test type: Other; Difference in percentage = 2.07, 95% CI 2-sided [-18.53 to 22.68] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: From dose 1 up to 28 days after end of study treatment (for OL1=maximum duration up to 16 weeks; for OL2= maximum duration up to 24 weeks and for DB=maximum duration up to 248 weeks)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both AE and non-SAE. OLPT1, OLPT2 and DBFAS analysis set was used.
Groups:
- Tofacitinib 5mg BID OL Part 1: Participants were administered tofacitinib 5 mg BID via the oral route and continued to receive a stable dose of corticosteroids during OL part 1.
- Tofacitinib 5mg BID OL Part 2: Participants who achieved sJIA ACR 50 response and maintained sJIA ACR 30 response for 4 weeks were administered tofacitinib 5 mg BID and tapering dose of CSs for participants treated with ˃0.2 mg/kg/day oral prednisone (or equivalent).
Arm/Group | Tofacitinib 5mg BID OL Part 1 | Tofacitinib 5mg BID OL Part 2 | Tofacitinib 5mg BID DB | Placebo DB
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/54 | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 7/100 | 0/54 | 0/28 | 2/31
Other Adverse Events (participants affected / at risk) | 33/100 | 15/54 | 23/28 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib 5mg BID OL Part 1 (N=100) | Tofacitinib 5mg BID OL Part 2 (N=54) | Tofacitinib 5mg BID DB (N=28) | Placebo DB (N=31)
Still's disease (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib 5mg BID OL Part 1 (N=100) | Tofacitinib 5mg BID OL Part 2 (N=54) | Tofacitinib 5mg BID DB (N=28) | Placebo DB (N=31)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (8) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 7 (11) | 3 (11) | 5 (19)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 6 (6) | 2 (8) | 4 (9) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (10)
Refraction disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Still's disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 8 (8) | 14 (14)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mycoplasma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03000439/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT03000439/SAP_001.pdf